CLINICAL TRIAL: NCT02003924
Title: PROSPER: A MULTINATIONAL, PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, EFFICACY AND SAFETY STUDY OF ENZALUTAMIDE IN PATIENTS WITH NONMETASTATIC CASTRATION-RESISTANT PROSTATE CANCER
Brief Title: Safety and Efficacy Study of Enzalutamide in Patients With Nonmetastatic Castration-Resistant Prostate Cancer
Acronym: PROSPER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDV3100-14; 2012-005665-12 (EudraCT Number); C3431005 (Other: Alias Study Number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Nonmetastatic Castration-Resistant Prostate Cancer; Prostate Cancer; Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Sham Comparator): Sugar pill manufactured to mimic enzalutamide 40 mg capsule
  Interventions: Drug: Placebo
- Enzalutamide (Experimental): 160 mg by mouth once daily
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — 160 mg by mouth once daily
  Other Names: MDV3100; Xtandi
  Arms: Enzalutamide
Drug: Placebo — Sugar pill to mimic enzalutamide
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of enzalutamide in patients with non metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, signet cell, or small cell features;
* Ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) agonist/antagonist or prior bilateral orchiectomy (medical or surgical castration);
* Testosterone ≤ 50 ng/dL (≤ 1.73 nmol/L) at screening;
* Progressive disease on androgen deprivation therapy at enrollment;
* PSA and the screening PSA assessed by the central laboratory (central PSA) should be ≥ 2 µg/L (2 ng/mL:
* PSA doubling time ≤ 10 months;
* No prior or present evidence of metastatic disease;
* Asymptomatic prostate cancer;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Estimated life expectancy ≥ 12 months.

Exclusion Criteria:

* Prior cytotoxic chemotherapy;
* Use of hormonal therapy or biologic therapy for prostate cancer (other than approved bone targeting agents and GnRH agonist/antagonist therapy) or use of an investigational agent within 4 weeks of randomization;
* Known or suspected brain metastasis or active leptomeningeal disease;
* History of another invasive cancer within 3 years of randomization;
* Absolute neutrophil count < 1000/μL, platelet count < 100,000/μL, or hemoglobin < 10 g/dL (6.2 mmol/L) at screening;
* Total bilirubin ≥ 1.5 times the upper limit of normal;
* Creatinine > 2 mg/dL (177 µmol/L) at screening;
* Albumin < 3.0 g/dL (30 g/L) at screening;
* History of seizure or any condition that may predispose to seizure;
* Clinically significant cardiovascular disease;
* Gastrointestinal disorder affecting absorption;
* Major surgery within 4 weeks of randomization;
* Hypersensitivity reaction to the active pharmaceutical ingredient or any of the capsule components, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene;
* Any concurrent disease, infection, or comorbid condition that interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of data, in the opinion of the investigator or medical monitor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1401 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2025-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (393):
- United States (37):
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Clark Urology Center, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Urology Associates of San Luis Obispo, a Medical Group, Inc, San Luis Obispo, California
  - Urology Associates, P.C., Englewood, Colorado
  - c/o Lynn Buchwalder, New Haven, Connecticut
  - C/O Thomas Ferencz, RPh, BCOP, Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Smilow Cancer Center at Yale New Haven-Hospital, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Urology of Indiana, LLC, Carmel, Indiana
  - First Urology, PSC, Jeffersonville, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Kansas City Urology Care, PA, Overland Park, Kansas
  - GU Research Network/ Wichita Urology Group, Wichita, Kansas
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - GU Research Network, Omaha, Nebraska
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Premier Medical Group of the Hudson Valley, Newburgh, New York
  - Duke University Medical Center, Cary, North Carolina
  - Carolina Urology Partners, PLLC, Charlotte, North Carolina
  - Carolina Urology Partners, PLLC, Gastonia, North Carolina
  - Gaston Medical Associates, Gastonia, North Carolina
  - Carolina Urology Partners, PLLC, Huntersville, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Lancaster Urology, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Dept. of Urologic Surgery, Nashville, Tennessee
  - Vanderbilt University Medical Center, The Urologic Clinic, Nashville, Tennessee
  - Urology San Antonio, San Antonio, Texas
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
- Argentina (9):
  - COIBA(Centro de Oncologia e Investigacion Buenos Aires), Berazategui, Buenos Aires
  - Centro Medico Austral(OMI), CABA, Buenos Aires
  - Centro de Urologia, CABA, Buenos Aires
  - Hospital Italiano de Buenos Aires, CABA, Buenos Aires
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Instituto De Oncologia De Rosario, Rosario, Santa Fe Province
  - Clinica Universidad Reina Fabiola, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Australia (38):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - The Border Cancer Hospital Dispensary, Albury, New South Wales
  - The Border Cancer Hospital, Albury, New South Wales
  - Sydney cancer centre, Concord, New South Wales
  - Epic pharmacy, Lismore, New South Wales
  - North Coast Cancer Institute, Lismore, New South Wales
  - Macquarie University Hospital, North Ryde, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Epic Pharmacy Port Macquarie base hospital, Port Macquarie, New South Wales
  - Mid North Coast Cancer Institute, Port Macquarie, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Australian Clinical Trials, Wahroonga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - River City Pharmacy - APHS, Auchenflower, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Integrated Clinical Oncology Network (ICON), South Brisbane, Queensland
  - Icon Cancer Care Southport, Southport, Queensland
  - Tasman Oncology Research Pty Ltd, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Cancer Care SA Pty Ltd, Kurralta Park, South Australia
  - Tenpharm Pty Ltd trading as EPIC Pharmacy Tennyson, Kurralta Park, South Australia
  - Box Hill Hospital (Eastern health), Box Hill, Victoria
  - Eastern Clinical Research Unit (Eastern Health), Box Hill, Victoria
  - Cabrini Hospital Brighton, Brighton, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Austin Hospital, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Cabrini Hospital- Education and Research Precinct, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Austria (6):
  - Krankenhaus Barmherzige Schwestern Linz, Abteilung Radiologie, Linz, Upper Austria
  - Krankenhaus Barmherzige Schwestern Linz, Abteilung Urologie, Linz, Upper Austria
  - St. Vincent's Hospital, PET - CT Center, Linz, Upper Austria
  - Isotopix, Ambulatorium fuer Nuklearmedizin, Vienna
  - Medizinische Universitaet Wien, Universitaetsklinik fuer Innere Medizin I, Vienna
  - Diagnosezentrum Meidling GesmbH, Vienna
- Belgium (5):
  - Algemeen Ziekenhuis Groeninge, Kortrijk, West-vlaanderen
  - Clinique Universitaire de Bruxelles Hopital Erasme, Brussels
  - Vzw Algemeen Ziekenhuis Maria Middelares, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege, Site du Sart-Tilman, Liège
- Brazil (17):
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Liga Paranaense de Combate ao cancer / Hospital Erasto Gaertner, Curitiba, Paraná
  - Instituto D'Or de Pesquisa e Ensino (IDOR), Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Hospital de Clínicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CLINIONCO - Clinica de Oncologia de Porto Alegre Ltda., Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Ciencias Medicas da UNICAMP, Campinas, São Paulo
  - Hospital Amaral Carvalho - Fundacao Dr. Amaral Carvalho, Jaú, São Paulo
  - Fundacao Dr. Amaral Carvalho, Jaú, São Paulo
  - Fundacao Dr.Amaral Carvalho, Jaú, São Paulo
  - Centro de Estudos e Pesquisas em Hematologia e Oncologia (CEPHO), Santo André, São Paulo
  - Hospital Israelita Albert Einstein, Sao Paulp, São Paulo
  - IAMSPE-Inst. de Assist. ao Servidor Publico Estadual, São Paulo, São Paulo
  - Hospital Universitario Pedro Ernesto - UERJ, Rio de Janeiro
  - Oncologia Rede D'Or, Rio de Janeiro
- Canada (16):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Manitoba Prostate Centre CancerCare Manitoba, Winnipeg, Manitoba
  - NS Health Authority, Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The Male/Female Health and Research Centre, Barrie, Ontario
  - McMaster Institute of Urology @ St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Urology Associates / Urologic Medical Research, Kitchener, Ontario
  - London Regional Cancer Program - Victoria Hospital, London Health Sciences Centre(LHSC), London, Ontario
  - Urology Reasearch - Victoria Hospital, London Health Sciences Centre(LHSC), London, Ontario
  - SunnyBrook Health Sciences Centre, Toronto, Ontario
  - University Health Network- Princess Margaret Cancer Centre, Toronto, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec, Québec, Quebec
- Chile (5):
  - Fundacion Arturo Lopez Perez, Santiago
  - Centro de Investigaciones Clinicas Vina del Mar, Santiago
  - Instituto Clinico Oncologico del Sur (ICOS), Temuco
  - Instituto Oncologico Ltda., Viña del Mar
  - Centro de Investigaciones Clinicas, Viña del Mar
- China (24):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Office of Hongqian Guo, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Qingdao Municipal Hospital (East Hospital), Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hosptial of Wenzhou Medical University, Wenzhou, Zhejiang
  - UNIMED Medical Institute Limited, Hong Kong
  - The Second Hospital of Tianjin Medical University, Tianjin
- Denmark (8):
  - Rigshospitalet 7521, Copenhagen, Norrebro
  - Copenhagen Prostate Cancer Center, Copenhagen, N
  - Aarhus University Hospital, Arhus N
  - Rigshospitalet, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense C
  - Vejle Sygehus, Vejle
- Finland (5):
  - Docrates Syopasairaala, Helsinki
  - Helsingin yliopistollinen keskussairaala, Meilahden sairaala, Helsinki
  - Oulun yliopistollinen sairaala, Oulu
  - Satakunnan keskussairaala, Pori
  - Tampereen yliopistollinen Sairaala, Tampere
- France (35):
  - Hopitaux Universitaires de Strasbourg - Hopital Civil, Strasbourg, Alsace
  - Centre Paul Strauss, Strasbourg, Bas-rhin
  - Clinique Sainte Anne, Strasbourg, Bas-rhin
  - Societe MIM, Clinique Sainte Anne, Strasbourg, Bas-rhin
  - Institut Curie, Paris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - Institut Gustave Roussy, Villejuif, VAL DE Marne
  - Institut de Cancerologie de l'Ouest - Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - Urologic Oncology Department- Institut Bergonie - Centre regional de Lutte contre le Cancer, Bordeaux
  - Cabinet de Radiologie, Brest
  - CHU Brest Hopital Morvan, Brest
  - Clinique pasteur Lancroze, Brest
  - Clinique Pasteur-Lanroze, Brest
  - CHRU de Brest, Brest
  - Hopital Pasteur, Colmar
  - Hopitaux Civils de Colmar, Colmar
  - Centre Regional de lutte Contre le Cancer Georges Francois Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Hopital Calude Huriez - CHU Lille, Lille
  - Centre de Medecine Nucleaire LUMEN, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - Hopital Nord, Marseille
  - ICM Val D'Aurelle, Montpellier
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Institut de Cancerologie de I'Ouest - Rene Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - IUCT-Oncopole, Toulouse
  - Clinique Pasteur - CIMOF, Toulouse
  - Clinique Pasteur- Service Imagerie et Radiologie, Toulouse
  - Clinique Pasteur, Toulouse
- Germany (14):
  - Universitatsmedizin Mannheim, Medizinische Fakultat Mannheim der Universitat Heidelberg, Mannheim, Baden-Wurttemberg
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - MVZ Zentrum fuer Diagnostische Radiologie und Nuklearmedizin Braunschweig GmbH, Braunschweig, Lower Saxony
  - Staedtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - Hannover Medical School, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - RWTH University Aachen, Aachen, North Rhine-Westphalia
  - Uniklinik der RWTH Aachen, Aachen, North Rhine-Westphalia
  - Clinic of Radiology, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Charite, Campus Benjamin Franklin, Berlin
  - Charite, Universitaetsmedizin Berlin, Berlin
  - Martini-Klinik am UKE GmbH, Hamburg
  - Diagnostikzentrum Esslingen, Kirchheim
- Greece (6):
  - University General Hospital of Heraklion, Urology Clinic, Heraklion, Crete
  - General Hospital of Athens"Korgialeneio-Benakeio EES".Urology Clinic, Athens
  - General Hospital of Athens "Alexandra", Therapeutic Clinic, Athens
  - University General Hospital of Larissa, Urology Department, Larissa
  - University General Hospital of Patras, Oncology Department, Internal Medicine Clinic, Pátrai
  - General Hospital" Papageorgiou",B' Univ.Urology Clinic, Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Italy (41):
  - Laboratorio Medicina Nucleare-Ospedale G.B. Morgagni-Pierantoni, Forlì, FC
  - Farmacia, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Medicina Nucleare, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Servizio di Radiologia, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Struttura Complessa di Oncologia, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - U.O. di Oncologia, Ospedale Civile Degli Infermi, Faenza (RA)
  - U.O. di Radiologia, Ospedale Civile degli Infermi, Faenza (RA)
  - U.O. di Oncologia, Ospedale Civile Umberto I, Lugo (RA)
  - U.O. di Radiologia, Ospedale Civile Umberto I, Lugo (RA)
  - Laboratorio Farmaci Antiblastici, Meldola (FC)
  - U.O. Oncologia Medica, Meldola (FC)
  - UO Radiologia, Meldola (FC)
  - Dipartimento di Radiologia, Ospedale San Raffaele, Milan
  - Servizio di Farmacia, Ospedale San Raffaele, Milan
  - U.O. di Medicina Nucleare e Centro PET, Ospedale San Raffaele, Milan
  - U.O. di Urologia, Ospedale San Raffaele, Milan
  - Farmacia Studi Clinici e Sperimentali, Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - S.C. di Oncologia Medica 1, Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - S.C. Diagnostica Radiologica 2, Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Divisione di Radiologia, Istituto Europeo di Oncologia, Milan
  - Reparto Oncologia Medica Urogenitale e Cervico Facciale, Istituto Europeo di Oncologia, Milan
  - Servizio Farmacia, Istituto Europeo di Oncologia, Milan
  - Farmacia Interna, Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Medicina Nucleare, Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Radiologia I, Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - U.O.S.C. di Oncologia Medica, A.O.R.N. "A. Cardarelli", Napoli
  - Farmacia Ospedaliera, AOU San Luigi Gonzaga, Orbassano (TO)
  - SCDU Oncologia Medica II Pad, AOU San Luigi Gonzaga, Orbassano (TO)
  - SCDU Radiodiagnostica, AOU San Luigi Gonzaga, Orbassano (TO)
  - SS Medicina Nucleare, AOU San Luigi Gonzaga, Orbassano (TO)
  - Farmacia, Istituto Oncologico Veneto (IOV), Padua
  - IRCCS - Istituto Oncologico Veneto (IOV), UOC Oncologia Medica 1, Padua
  - Medicina Nucleare, Istituto Oncologico Veneto (IOV), Padua
  - UOC Radiodiagnostica Oncologica, Istituto Oncologico Veneto (IOV), Padua
  - Dipartimento di Onco-Ematologia Ospedale Santa Maria delle Croci, Ravenna
  - Servizio di Farmacia, AUSL di Ravenna, Ravenna
  - Servizio di Radiologia, AUSL di Ravenna, Ravenna
  - Azienda Ospedaliera S. Camillo Forlanini, UOC per il governo clinico in Oncologia Medica, Roma
  - U.O. di Oncologia Medica, Ospedale Santa Chiara, Trento
  - U.O. Farmacia, Ospedale Santa Chiara, Trento
  - U.O. Radiologia, Ospedale Santa Chiara, Trento
- Malaysia (5):
  - Universiti Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
  - Subang Jaya Medical Centre Sdn. Bhd., Subang Jaya, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Netherlands (6):
  - Maastricht University Medical Centre, Maastricht, AZ
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Netherlands Cancer Institute, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - University Medical Center Groningen, Groningen
  - Radboud University Nijmegen Medical Centre, Nijmegen
- New Zealand (4):
  - Canterbury District Health Board, Christchurch, Canterbury
  - Palmerston North Hospital, Palmerston North, Manawatu
  - Waikato Urology Research LTD, Hamilton, Waikato Region
  - Cancer and Blood Research, Auckland
- Poland (9):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - UROMEDYK, Poradnia Urologiczna, Kielce
  - Malopolskie Centrum Medyczne s.c., Krakow
  - Wojewodzki Szpital Specjalistyczny im. Stefana Kardynala Wyszynskiego SPZOZ, Lublin
  - Wojewodzki Szpital Specjalistyczny im. Janusza. Korczaka, Słupsk
  - Profesorskie Centrum Medyczne Optimum, Wroclaw
  - Centrum Medyczne Melita Medical, Wroclaw
  - Wro Medica, Wroclaw
  - Lexmedica, Wroclaw
- Russia (7):
  - Federal State Budgetary Institution "N.N. Blokhin Russian Cancer Research Center", Moscow
  - P. Hertsen Moscow Oncology Research Institute - branch of the National Medical Research, Moscow
  - State Budgetary Healthcare Institution City Multifield Hospital No.2, Saint Petersburg
  - SBEI HPE "First Pavlov State Medical University of St. Petersburg" of, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "Hospital for Veterans of War", Saint Petersburg
  - SBHI "Saint-Petersburg clinical scientific, Saint Petersburg
  - SBEI of HPE "Bashkir State Medical University" of MoH of the RF, Ufa
- Serbia (4):
  - Clinical Center Of Serbia, Clinic of Urology, Belgrade
  - Clinical Center "Dr Dragisa Misovic -Dedinje", Clinic of Urology, Belgrade
  - Clinical Center "Bezanijska Kosa", Department of Urology, Belgrade
  - Clinical Center Zemun, Belgrade
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- Slovakia (19):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Institut nuklearnej a molekularnej mediciny, Banská Bystrica
  - Bratislavske radiodiagnosticke centrum, a.s., Bratislava
  - CUIMED, s.r.o., Urologicka ambulancia, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - Institut nuklearnej a molekularnej mediciny, Košice
  - Univerzitna nemocnica Martin, Martin
  - IZOTOPCENTRUM, s.r.o., Nitra
  - Jessenius-diagnosticke centrum, a.s., Nitra
  - UROEXAM spol. s r.o. urologicka ambulancia, Nitra
  - Alfamedis, s.r.o., Prešov
  - MILAB s.r.o., UROCENTRUM, Prešov
  - Vivamed, s.r.o, Prešov
  - UVN SNP - FN Ruzomberok, Pracovisko Nuklearnej mediciny CCSR, Ružomberok
  - Fakultna nemocnica s Poliklinikou Skalica a.s, Skalica
  - GAMMALAB, spol. s.r.o., Oddelenie nuklearnej mediciny, Trnava
  - GAMMALAB, spol.s.r.o., Oddelenie nuklearnej mediciny, Trnava
  - KK MED s.r.o., Žilina
  - Fakultna nemocnica s poliklinikou Zilina, Urologicke oddelenie, Žilina
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (14):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitari Son Espases,, Palma de Mallorca, Balearic Islands
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - ALTAHIA. Xarxa Assistencial Universitaria de Manresa, Manresa, Barcelona
  - Hospital Universitario Parc Tauli, Sabadell, Barcelona
  - ICO Girona-Hospital Universitari de Girona Dr. Josep Trueta, Girona, Catalonia
  - Hospital de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Del Mar, Barcelona
  - Cetir Centre Medic, S.L., Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 de octubre, Madrid
- Sweden (8):
  - Urologmottagningen, Gothenburg
  - Diagnostiskt centrum for bild- och funktionsmedicin, Malmo
  - Urologiska Kliniken, Malmo
  - Apoteket AB Kliniska Provningar Molnlycke, Mölnlycke
  - Urologiska Kliniken, Örebro
  - Karolinska Universitetssjukhuset, Solna
  - Urologmottagningen, Stockholm
  - Urologkliniken, Umeå
- Taiwan (11):
  - Chang Gung Medical Fundation, Chiayi Branch(Chiayi Chang Gung Memorial Hospital), Chiayi County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Medical Fundation,Kaohsiung (Kaohsiung Chang Gung Memorial Hospital), Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung Branch (Keelung Chang Gung Memorial Hospital), Keelung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Centre, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital at Linkuo, Taoyuan
- Thailand (4):
  - Songklanagarind hospital, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Muang, Chiang Mai
  - King Chulalongkorn Memorial Hospital, Chulalongkorn University, Bangkok
  - Rajavithi Hospital, Bangkok
- Turkey (Türkiye) (5):
  - Cukurova Universitesi Tip Fakultesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Izmir Bozyaka Egitim Arastirma Hastanesi, Izmir
  - Celal Bayar Universitesi Tip Fakultesi, Manisa
- Ukraine (6):
  - RCI Chernivtsi Regional Clinical Hospital, Chernivtsi
  - CI I.I. Mechnikov DRCH Dept of Urology #2, Dnipropetrovsk
  - CHI V.I.Shapoval RCC of Urology and Nephrology, Dep. Of Urology#4, Kharkiv
  - CNE Kyiv City Clinical Hospital #3 of Ex Body of KCC (Kyiv CSA), Department of Urology, Kyiv
  - Central City Clinical Hospital, City Oncological Center, Uzhhorod
  - CI Zaporizhzhia Regional Clinical Hospital, Dep. Of Urology,, Zaporizhzhia
- United Kingdom (12):
  - East and North Hertfordshire NHS Trust, Northwood, Middlesex
  - Belfast Health and Social Care Trust, Belfast, Northern Ireland
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, TYNE and WEAR
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University College Hospitals NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hussain M, Sternberg CN, Efstathiou E, Fizazi K, Shen Q, Lin X, Sugg J, Steinberg J, Noerby B, De Giorgi U, Shore ND, Saad F. Nadir Prostate-specific Antigen as an Independent Predictor of Survival Outcomes: A Post Hoc Analysis of the PROSPER Randomized Clinical Trial. J Urol. 2023 Mar;209(3):532-539. doi: 10.1097/JU.0000000000003084. Epub 2023 Feb 9. PMID 36756959
- [Derived] De Giorgi U, Hussain M, Shore N, Fizazi K, Tombal B, Penson D, Saad F, Efstathiou E, Madziarska K, Steinberg J, Sugg J, Lin X, Shen Q, Sternberg CN. Which traits affect how long patients with advanced prostate cancer live when treated with enzalutamide? Future Oncol. 2022 Nov;18(35):3867-3874. doi: 10.2217/fon-2022-0661. Epub 2022 Oct 13. PMID 36226865
- [Derived] Cella D, Ganguli A, Turnbull J, Rohay J, Morlock R. US Population Reference Values for Health-Related Quality of Life Questionnaires Based on Demographics of Patients with Prostate Cancer. Adv Ther. 2022 Aug;39(8):3696-3710. doi: 10.1007/s12325-022-02204-3. Epub 2022 Jun 22. PMID 35731340
- [Derived] Joshua AM, Armstrong A, Crumbaker M, Scher HI, de Bono J, Tombal B, Hussain M, Sternberg CN, Gillessen S, Carles J, Fizazi K, Lin P, Duggan W, Sugg J, Russell D, Beer TM. Statin and metformin use and outcomes in patients with castration-resistant prostate cancer treated with enzalutamide: A meta-analysis of AFFIRM, PREVAIL and PROSPER. Eur J Cancer. 2022 Jul;170:285-295. doi: 10.1016/j.ejca.2022.04.005. Epub 2022 May 26. PMID 35643841
- [Derived] De Giorgi U, Hussain M, Shore N, Fizazi K, Tombal B, Penson D, Saad F, Efstathiou E, Madziarska K, Steinberg J, Sugg J, Lin X, Shen Q, Sternberg CN. Consistent survival benefit of enzalutamide plus androgen deprivation therapy in men with nonmetastatic castration-resistant prostate cancer: PROSPER subgroup analysis by age and region. Eur J Cancer. 2021 Dec;159:237-246. doi: 10.1016/j.ejca.2021.10.015. Epub 2021 Nov 14. PMID 34784577
- [Derived] Saad F, Sternberg CN, Efstathiou E, Fizazi K, Modelska K, Lin X, Sugg J, Steinberg J, Noerby B, Shore ND, Hussain M. Prostate-specific Antigen Progression in Enzalutamide-treated Men with Nonmetastatic Castration-resistant Prostate Cancer: Any Rise in Prostate-specific Antigen May Require Closer Monitoring. Eur Urol. 2020 Dec;78(6):847-853. doi: 10.1016/j.eururo.2020.08.025. Epub 2020 Oct 1. PMID 33010985
- [Derived] Sternberg CN, Fizazi K, Saad F, Shore ND, De Giorgi U, Penson DF, Ferreira U, Efstathiou E, Madziarska K, Kolinsky MP, Cubero DIG, Noerby B, Zohren F, Lin X, Modelska K, Sugg J, Steinberg J, Hussain M; PROSPER Investigators. Enzalutamide and Survival in Nonmetastatic, Castration-Resistant Prostate Cancer. N Engl J Med. 2020 Jun 4;382(23):2197-2206. doi: 10.1056/NEJMoa2003892. Epub 2020 May 29. PMID 32469184
- [Derived] Tombal B, Saad F, Penson D, Hussain M, Sternberg CN, Morlock R, Ramaswamy K, Ivanescu C, Attard G. Patient-reported outcomes following enzalutamide or placebo in men with non-metastatic, castration-resistant prostate cancer (PROSPER): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2019 Apr;20(4):556-569. doi: 10.1016/S1470-2045(18)30898-2. Epub 2019 Feb 12. PMID 30770294
- [Derived] Hussain M, Fizazi K, Saad F, Rathenborg P, Shore N, Ferreira U, Ivashchenko P, Demirhan E, Modelska K, Phung D, Krivoshik A, Sternberg CN. Enzalutamide in Men with Nonmetastatic, Castration-Resistant Prostate Cancer. N Engl J Med. 2018 Jun 28;378(26):2465-2474. doi: 10.1056/NEJMoa1800536. PMID 29949494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 254 sites in 32 countries.
Pre-assignment Details: A protocol amendment was implemented to unblind all participants and those who were previously treated with placebo had an opportunity to receive open-label access to enzalutamide at the discretion of the investigator.
Groups:
- Enzalutamide 160 mg: Participants received 4 capsules of Enzalutamide 40 mg each (total dose 160 mg per day) orally, once daily in double-blind and open-label phase (up to a maximum of 68.8 months) until radiographic progression. Participants after last dose of study drug, were followed up for safety up to 30 days, and were long term followed up (for survival status and new prostate cancer therapies) from last dose to the death date or last known survival date.
- Placebo: Participants received 4 capsules of placebo (matched to Enzalutamide) orally, once daily in double blind phase (up to a maximum of 51.3 months) until radiographic progression. Participants were given an opportunity to switch to open-label enzalutamide after completion of double blind phase. Participants after last dose of study drug, were followed up for safety up to 30 days and were long term followed up (for survival status and new prostate cancer therapies) to the death date or last known survival date.
- Placebo Participants Crossover to Enzalutamide 160 mg: Participants who received placebo in double-blind phase and who agreed to proceed to open-label phase, received 4 capsules of Enzalutamide 40 mg each (total dose of 160 mg per day), orally once daily (up to a maximum of 18.8 months) until radiographic progression. Participants after last dose of study drug, were followed up for safety up to 30 days and were long term followed up (for survival status and new prostate cancer therapies) to the death date or last known survival date.
Period: Double-blind Phase
Arm/Group | Enzalutamide 160 mg | Placebo | Placebo Participants Crossover to Enzalutamide 160 mg
Started | 933 | 468 | 0
Treated | 930 | 465 | 0
Completed | 478 | 87 | 0
Not Completed | 455 | 381 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Withdrawal Consent to Continue Treatment | 71 | 47 | 0
Not completed — Disease Progression | 229 | 247 | 0
Not completed — Adverse Event | 120 | 31 | 0
Not completed — Randomized But not Treated | 3 | 3 | 0
Not completed — Other | 29 | 50 | 0
Period: Open-label Phase
Arm/Group | Enzalutamide 160 mg | Placebo | Placebo Participants Crossover to Enzalutamide 160 mg
Started | 478 | 0 (Participants were offered to switch from double blind placebo to open label Enzalutamide.) | 87 (Participants previously treated with placebo, switched to receive open label Enzalutamide.)
Treated | 478 | 0 | 87
Completed | 378 | 0 | 70
Not Completed | 100 | 0 | 17
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal Consent to Continue Treatment | 9 | 0 | 1
Not completed — Disease Progression | 59 | 0 | 5
Not completed — Adverse Event | 25 | 0 | 10
Not completed — Other | 7 | 0 | 0
Period: Long-term Follow-up Phase
Arm/Group | Enzalutamide 160 mg | Placebo | Placebo Participants Crossover to Enzalutamide 160 mg
Started | 933 (Participants followed up after discontinuing study drug in either double blind or open label phase.) | 381 (Participants were followed up after study drug discontinuation in double blind phase.) | 87 (Participants were followed up after study drug discontinuation in open label phase.)
Completed | 566 | 144 | 80
Not Completed | 367 | 237 | 7
Not completed — Death | 288 | 174 | 4
Not completed — Lost to Follow-up | 8 | 6 | 1
Not completed — Withdrew Consent to Be Followed | 66 | 55 | 1
Not completed — Other | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all participants randomly assigned to study treatment and was based on randomized treatment assignment regardless of whether or not treatment was administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzalutamide 160 mg | Placebo | Total
Number analyzed (Participants) | 933 | 468 | 1401
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (7.83) | 72.9 (7.63) | 73.5 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 933 | 468 | 1401
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 142 | 88 | 230
  Black or African American | 21 | 10 | 31
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  White | 671 | 320 | 991
  Multiple | 4 | 4 | 8
  Other | 15 | 5 | 20
  Missing | 77 | 39 | 116

OUTCOME MEASURES:

1. Primary Outcome: Metastasis Free Survival (MFS)
Description: MFS:time from randomization to first date of radiographic progression (RP) (by Blinded independent central radiology review [BICR]) at any time or death within 112 days of treatment discontinuation without evidence of RP.RP for bone disease:appearance of 1 or more metastatic lesions on bone scan.RP for soft tissue disease:per Response Evaluation Criteria in Solid Tumors,[RECIST 1.1])-at least a 20 percent (%) increase in the sum of diameters of target lesions,taking as reference the smallest sum on study (includes the baseline sum if smallest on study).Participants who did not have MFS event at the time of analysis data cut-off (28 June 2017) were censored at date of last assessment showing no objective evidence of RP prior to skeletal-related event or two or more consecutive missed tumor assessments. Participants who were randomized but later confirmed to have metastatic disease before randomization were censored on date of randomization. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization until radiographic progression at any time, or death within 112 days of treatment discontinuation, whichever occurred first (until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | 36.6 [33.1 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events. | 14.7 [14.2 to 15.0]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — P-value was based on stratified log-rank test by prostate-specific antigen (PSA) doubling time (< 6 months, >= 6 months) and prior or concurrent use of a bone targeting agent (yes, no). Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.292, 95% CI 2-sided [0.241 to 0.352] — HR was based on a Cox regression model (with treatment as the only covariate) stratified by factors defined above, and was relative to placebo with < 1 favoring Enzalutamide

2. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as the time from randomization to the date of first PSA value demonstrating progression, which was subsequently confirmed. For participants with PSA decline at Week 17, PSA progression was defined according to Prostate Cancer Working Group 2 (PCWG2) guidelines as the date that a 25% or greater increase and an absolute increase of 2 nanograms per milliliter (ng/mL) above the nadir (or baseline for participants with no PSA decline by Week 17) was documented, which was confirmed by a second consecutive value obtained at least 3 weeks or later. Participants without confirmed PSA progression at the time of analysis were right censored at the date of last PSA assessment before the analysis data cut-off date for the purposes of analysis. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization until first PSA progression (until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: The ITT population was defined as all participants randomly assigned to study treatment and was based on randomized treatment assignment regardless of whether or not treatment was administered.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | 37.2 [33.1 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events. | 3.9 [3.8 to 4.0]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg vs Placebo; To maintain the family-wise 2-sided type I error rate at 0.05, a parallel testing strategy between OS (with allocated type I error rate 0.03) and remaining key secondary endpoints (time to PSA progression and time to first use of new antineoplastic therapy with allocated type I error rate 0.02) was performed. Testing was performed only if the primary endpoint was statistically significant; Test type: Superiority; p < 0.0001, Log Rank — P-value was based on a stratified log-rank test by PSA doubling time (< 6 months, >= 6 months) and prior or concurrent use of a bone targeting agent (yes, no) as per IXRS. Threshold for significance at 0.02 level; Hazard Ratio (HR) = 0.066, 95% CI 2-sided [0.054 to 0.081] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to First Use of New Antineoplastic Therapy
Description: Time to first use of new antineoplastic therapy was defined as the time from randomization to first use of new antineoplastic for prostate cancer. Participants not starting treatment with a new antineoplastic therapy at the time of analysis were right censored at the date of last assessment before the analysis data cutoff date for the purposes of analysis. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization until first use of new antineoplastic therapy(until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | 39.6 [37.7 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events. | 17.7 [16.2 to 19.7]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg vs Placebo; To maintain the family-wise 2-sided type I error rate at 0.05, a parallel testing strategy between OS (with allocated type I error rate 0.03) and remaining key secondary endpoints (time to PSA progression and time to first use of new antineoplastic therapy with allocated type I error rate 0.02) was performed. Testing was performed only if the previous endpoint was statistically significant; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.208, 95% CI 2-sided [0.168 to 0.258] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time (in months) from randomization to death from any cause. For participants who were alive at the time of the analysis data cutoff, OS time was censored at the last date the participant was known to be alive or analysis data cutoff date, whichever was earlier. Participants with no post baseline survival information were censored on the date of randomization. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization until death (up to a maximum of 68.8 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | 67.0 [64.0 to NA] — Lower limit for 95% CI could not be estimated because there were insufficient number of participants with event. | 56.3 [54.4 to 63.0]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg vs Placebo; To maintain family-wise 2-sided type I error rate at 0.05,parallel testing strategy between OS(with allocated type I error rate 0.03)and remaining key secondary endpoints(time to PSA progression and time to first use of new antineoplastic therapy with allocated type I error rate 0.02)was performed.OS tested at error rate 0.05 when both time to PSA progression and time to first use of new antineoplastic therapy were significant. When either failed to show significance.OS was tested at error 0.03; Test type: Superiority; p = 0.0011, Log Rank — P-value was based on a stratified log-rank test by PSA doubling time (< 6 months, >= 6 months) and prior or concurrent use of a bone targeting agent (yes, no) as per interactive voice/web recognition system (IXRS); Hazard Ratio (HR) = 0.734, 95% CI 2-sided [0.608 to 0.885] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Pain Progression
Description: Pain was assessed using the score from the Brief Pain Inventory-Short Form (BPI-SF) question 3: "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the last 24 hours." Time to this event was defined as the time from randomization to onset of pain progression, where pain progression was defined as a 2-point or more increase from baseline in the question 3 score. Participants without observed pain progression at the time of analysis were right censored at the date of last pain assessment for the purposes of analysis. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization until onset of pain progression (until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | 18.5 [17.0 to 22.1] | 18.4 [14.8 to 22.1]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg vs Placebo; Test type: Superiority; p = 0.6534, Log Rank — P-value was based on a stratified log-rank test by PSA doubling time (< 6 months, >= 6 months) and prior or concurrent use of a bone targeting agent (yes, no) as per IXRS; Hazard Ratio (HR) = 0.959, 95% CI 2-sided [0.801 to 1.149] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to First Use of Cytotoxic Chemotherapy
Description: Time to first use of cytotoxic chemotherapy was defined as the time from randomization to the first use of cytotoxic chemotherapy for prostate cancer. Participants not starting treatment with a cytotoxic chemotherapy for prostate cancer at the time of analysis were right censored at the date of last assessment before the analysis data cutoff date for the purposes of analysis. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization up to the first use of cytotoxic chemotherapy (until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | NA [38.1 to NA] — The median and upper limit of the 95% CI was not estimable due to the small number of events. | 39.7 [38.9 to 41.3]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 5, analysis 1]; Hazard Ratio (HR) = 0.378, 95% CI 2-sided [0.282 to 0.507] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Chemotherapy-Free Disease Specific Survival
Description: Chemotherapy-free disease-specific survival was defined as the time from randomization to first use of cytotoxic chemotherapy for prostate cancer or death due to prostate cancer as assessed by the investigator. Participants not starting treatment with a cytotoxic chemotherapy or not known to have died due to prostate cancer at the time of analysis were right censored at the date of last assessment before the analysis data cutoff date for the purposes of analysis. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization up to first use of cytotoxic chemotherapy for prostate cancer or death due to prostate cancer (until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | 39.6 [37.7 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events. | 38.9 [30.9 to 41.3]

8. Secondary Outcome: Chemotherapy-Free Survival
Description: Chemotherapy-free survival was defined as the time from randomization to first use of cytotoxic chemotherapy for prostate cancer or death due to any cause. Participants not starting treatment with a cytotoxic chemotherapy or not known to have died at the time of analysis were censored at the date of last assessment before the analysis data cutoff date for the purposes of analysis. Analysis was based on Kaplan-Meier estimates.
Time Frame: From randomization up to first use of cytotoxic chemotherapy for prostate cancer or death due to any cause (until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
months | 38.1 [37.7 to NA] — The upper limit of the 95% CI was not estimable due to the small number of events. | 34.0 [30.3 to 39.7]

9. Secondary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: PSA response was calculated at each visit as a decline from baseline in PSA (ng/mL) to the maximal PSA response with thresholds at 50% and 90%. Additionally, PSA response was assessed as a decline to undetectable levels, where undetectable level was defined as below the limit of quantification of the centrally assessed PSA results (the lower limit of quantification was 0.02 ng/mL). PSA response was confirmed by a second consecutive value at least 3 weeks later.
Time Frame: as for outcome 2
Population: The ITT population was defined as all participants randomly assigned to study treatment and was based on randomized treatment assignment regardless of whether or not treatment was administered. Here, 'Overall number of participants analyzed' = participants with baseline and at least one post-baseline PSA assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
percentage of participants
  Decrease from Baseline >= 50% | 76.3 [73.5 to 79.0] | 2.4 [1.2 to 4.2]
  Decrease from Baseline >= 90% | 55.9 [52.7 to 59.2] | 0.4 [0.1 to 1.5]
  Decrease to Undetectable Level | 9.6 [7.8 to 11.7] | 0 [0 to 0.8]
Statistical Analysis 1: Comparison: Enzalutamide 160 mg vs Placebo; Decrease from Baseline >= 50%; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was based on a Cochran-Mantel-Haenszel mean score test stratified by PSA doubling time (<6 months, >= 6 months) and prior concurrent use of a bone targeting agent (yes, no) as per IXRS; Difference in Response Rate = 73.96, 95% CI 2-sided [70.91 to 77.02]
Statistical Analysis 2: Comparison: Enzalutamide 160 mg vs Placebo; Decrease from Baseline >= 90%; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Difference in Response Rate = 55.52, 95% CI 2-sided [52.28 to 58.76]
Statistical Analysis 3: Comparison: Enzalutamide 160 mg vs Placebo; Decrease to Undetectable Level; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 9, analysis 1]; Difference in Response Rate = 9.65, 95% CI 2-sided [7.75 to 11.54]

10. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by Functional Assessment of Cancer Therapy-Prostate (FACT-P) Global Score
Description: The FACT-P questionnaire is a multidimensional, self-reported quality of life instrument consisting of 27 core items that assess participant function in 4 domains: physical, social/family, emotional, functional well-being, and supplemented by 12 site-specific items to assess prostate-related symptoms. Each item was rated on a 0 to 4 Likert-type scale, and then combined to produce subscale scores for each domain, as well as a global quality of life score which ranged from 0 to 156 where higher scores represented better quality of life.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: The ITT population was defined as all participants randomly assigned to study treatment and was based on randomized treatment assignment regardless of whether or not treatment was administered. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
units on a scale
  Baseline: number analyzed (Participants) | 887 | 439
  Baseline | 119.5 (17.75) | 120.8 (16.73)
  Change at Week 17: number analyzed (Participants) | 815 | 403
  Change at Week 17 | -4.0 (14.03) | -3.0 (13.87)
  Change at Week 33: number analyzed (Participants) | 718 | 329
  Change at Week 33 | -4.6 (14.82) | -3.5 (13.74)
  Change at Week 49: number analyzed (Participants) | 621 | 239
  Change at Week 49 | -3.9 (14.70) | -5.0 (15.71)
  Change at Week 65: number analyzed (Participants) | 522 | 183
  Change at Week 65 | -4.0 (15.84) | -5.7 (15.04)
  Change at Week 81: number analyzed (Participants) | 427 | 139
  Change at Week 81 | -4.1 (15.01) | -7.5 (16.42)
  Change at Week 97: number analyzed (Participants) | 354 | 90
  Change at Week 97 | -4.9 (15.31) | -5.9 (15.80)
  Change at Week 113: number analyzed (Participants) | 264 | 68
  Change at Week 113 | -5.5 (16.07) | -5.8 (13.16)
  Change at Week 129: number analyzed (Participants) | 186 | 37
  Change at Week 129 | -6.3 (17.33) | -8.1 (13.99)
  Change at Week 145: number analyzed (Participants) | 109 | 17
  Change at Week 145 | -5.5 (18.75) | -9.8 (15.47)
  Change at Week 161: number analyzed (Participants) | 38 | 6
  Change at Week 161 | -8.9 (19.88) | -7.0 (10.95)
  Change at Week 177: number analyzed (Participants) | 5 | 1
  Change at Week 177 | -4.8 (13.19) | -5.0

11. Secondary Outcome: Number of Participants With European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Mobility Domain Score
Description: EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Number of participants with various responses to the mobility questionnaire are reported.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: The ITT population was defined as all participants randomly assigned to study treatment and was based on randomized treatment assignment regardless of whether or not treatment was administered. Here, 'Number analyzed' = Participants evaluable for this outcome measure for specified categories.
Measure: Number; unit: participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
participants
  Baseline-No problem in walking: number analyzed (Participants) | 884 | 439
  Baseline-No problem in walking | 578 | 298
  Baseline-slight problem in walking: number analyzed (Participants) | 884 | 439
  Baseline-slight problem in walking | 183 | 100
  Baseline-moderate problem in walking: number analyzed (Participants) | 884 | 439
  Baseline-moderate problem in walking | 100 | 33
  Baseline-severe problem in walking: number analyzed (Participants) | 884 | 439
  Baseline-severe problem in walking | 21 | 7
  Baseline-unable to walk: number analyzed (Participants) | 884 | 439
  Baseline-unable to walk | 2 | 1
  Week 17-no problem in walking: number analyzed (Participants) | 840 | 419
  Week 17-no problem in walking | 526 | 274
  Week 17-slight problem in walking: number analyzed (Participants) | 840 | 419
  Week 17-slight problem in walking | 190 | 88
  Week 17-moderate problem in walking: number analyzed (Participants) | 840 | 419
  Week 17-moderate problem in walking | 87 | 50
  Week 17-severe problem in walking: number analyzed (Participants) | 840 | 419
  Week 17-severe problem in walking | 32 | 6
  Week 17-unable to walk: number analyzed (Participants) | 840 | 419
  Week 17-unable to walk | 5 | 1
  Week 33-no problem in walking: number analyzed (Participants) | 738 | 342
  Week 33-no problem in walking | 431 | 223
  Week 33-slight problem in walking: number analyzed (Participants) | 738 | 342
  Week 33-slight problem in walking | 162 | 85
  Week 33-moderate problem in walking: number analyzed (Participants) | 738 | 342
  Week 33-moderate problem in walking | 103 | 24
  Week 33-severe problem in walking: number analyzed (Participants) | 738 | 342
  Week 33-severe problem in walking | 36 | 10
  Week 33-unable to walk: number analyzed (Participants) | 738 | 342
  Week 33-unable to walk | 6 | 0
  Week 49-no problem in walking: number analyzed (Participants) | 635 | 250
  Week 49-no problem in walking | 362 | 156
  Week 49-slight problem in walking: number analyzed (Participants) | 635 | 250
  Week 49-slight problem in walking | 158 | 57
  Week 49-moderate problem in walking: number analyzed (Participants) | 635 | 250
  Week 49-moderate problem in walking | 86 | 27
  Week 49-severe problem in walking: number analyzed (Participants) | 635 | 250
  Week 49-severe problem in walking | 25 | 8
  Week 49-unable to walk: number analyzed (Participants) | 635 | 250
  Week 49-unable to walk | 4 | 2
  Week 65-no problem in walking: number analyzed (Participants) | 536 | 193
  Week 65-no problem in walking | 319 | 121
  Week 65-slight problem in walking: number analyzed (Participants) | 536 | 193
  Week 65-slight problem in walking | 109 | 44
  Week 65-moderate problem in walking: number analyzed (Participants) | 536 | 193
  Week 65-moderate problem in walking | 75 | 22
  Week 65-severe problem in walking: number analyzed (Participants) | 536 | 193
  Week 65-severe problem in walking | 29 | 6
  Week 65-unable to walk: number analyzed (Participants) | 536 | 193
  Week 65-unable to walk | 4 | 0
  Week 81-no problem in walking: number analyzed (Participants) | 435 | 148
  Week 81-no problem in walking | 236 | 88
  Week 81-slight problem in walking: number analyzed (Participants) | 435 | 148
  Week 81-slight problem in walking | 111 | 39
  Week 81-moderate problem in walking: number analyzed (Participants) | 435 | 148
  Week 81-moderate problem in walking | 61 | 15
  Week 81-severe problem in walking: number analyzed (Participants) | 435 | 148
  Week 81-severe problem in walking | 26 | 4
  Week 81-unable to walk: number analyzed (Participants) | 435 | 148
  Week 81-unable to walk | 1 | 2
  Week 97-no problem in walking: number analyzed (Participants) | 365 | 95
  Week 97-no problem in walking | 189 | 59
  Week 97-slight problem in walking: number analyzed (Participants) | 365 | 95
  Week 97-slight problem in walking | 94 | 24
  Week 97-moderate problem in walking: number analyzed (Participants) | 365 | 95
  Week 97-moderate problem in walking | 54 | 8
  Week 97-severe problem in walking: number analyzed (Participants) | 365 | 95
  Week 97-severe problem in walking | 22 | 4
  Week 97-unable to walk: number analyzed (Participants) | 365 | 95
  Week 97-unable to walk | 6 | 0
  Week 113-no problem in walking: number analyzed (Participants) | 275 | 73
  Week 113-no problem in walking | 140 | 45
  Week 113-slight problem in walking: number analyzed (Participants) | 275 | 73
  Week 113-slight problem in walking | 76 | 14
  Week 113-moderate problem in walking: number analyzed (Participants) | 275 | 73
  Week 113-moderate problem in walking | 41 | 11
  Week 113-severe problem in walking: number analyzed (Participants) | 275 | 73
  Week 113-severe problem in walking | 14 | 2
  Week 113-unable to walk: number analyzed (Participants) | 275 | 73
  Week 113-unable to walk | 4 | 1
  Week 129-no problem in walking: number analyzed (Participants) | 193 | 41
  Week 129-no problem in walking | 94 | 26
  Week 129-slight problem in walking: number analyzed (Participants) | 193 | 41
  Week 129-slight problem in walking | 48 | 9
  Week 129-moderate problem in walking: number analyzed (Participants) | 193 | 41
  Week 129-moderate problem in walking | 36 | 5
  Week 129-severe problem in walking: number analyzed (Participants) | 193 | 41
  Week 129-severe problem in walking | 15 | 1
  Week 129-unable to walk: number analyzed (Participants) | 193 | 41
  Week 129-unable to walk | 0 | 0
  Week 145-no problem in walking: number analyzed (Participants) | 116 | 21
  Week 145-no problem in walking | 56 | 13
  Week 145-slight problem in walking: number analyzed (Participants) | 116 | 21
  Week 145-slight problem in walking | 35 | 5
  Week 145-moderate problem in walking: number analyzed (Participants) | 116 | 21
  Week 145-moderate problem in walking | 18 | 2
  Week 145-severe problem in walking: number analyzed (Participants) | 116 | 21
  Week 145-severe problem in walking | 7 | 1
  Week 145-unable to walk: number analyzed (Participants) | 116 | 21
  Week 145-unable to walk | 0 | 0
  Week 161-no problem in walking: number analyzed (Participants) | 40 | 8
  Week 161-no problem in walking | 22 | 2
  Week 161-slight problem in walking: number analyzed (Participants) | 40 | 8
  Week 161-slight problem in walking | 7 | 5
  Week 161-moderate problem in walking: number analyzed (Participants) | 40 | 8
  Week 161-moderate problem in walking | 6 | 1
  Week 161-severe problem in walking: number analyzed (Participants) | 40 | 8
  Week 161-severe problem in walking | 5 | 0
  Week 161-unable to walk: number analyzed (Participants) | 40 | 8
  Week 161-unable to walk | 0 | 0
  Week 177-no problem in walking: number analyzed (Participants) | 6 | 1
  Week 177-no problem in walking | 3 | 0
  Week 177-slight problem in walking: number analyzed (Participants) | 6 | 1
  Week 177-slight problem in walking | 2 | 1
  Week 177-moderate problem in walking: number analyzed (Participants) | 6 | 1
  Week 177-moderate problem in walking | 1 | 0
  Week 177-severe problem in walking: number analyzed (Participants) | 6 | 1
  Week 177-severe problem in walking | 0 | 0
  Week 177-unable to walk: number analyzed (Participants) | 6 | 1
  Week 177-unable to walk | 0 | 0

12. Secondary Outcome: Number of Participants With European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Self-Care Domain Score
Description: EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ VAS. EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Number of participants with various responses to the self-care questionnaire are reported.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
participants
  Baseline:no problems washing or dressing: number analyzed (Participants) | 884 | 439
  Baseline:no problems washing or dressing | 805 | 415
  Baseline:slight problems washing or dressing: number analyzed (Participants) | 884 | 439
  Baseline:slight problems washing or dressing | 51 | 23
  Baseline:moderate problems washing or dressing: number analyzed (Participants) | 884 | 439
  Baseline:moderate problems washing or dressing | 22 | 1
  Baseline:severe problems washing or dressing: number analyzed (Participants) | 884 | 439
  Baseline:severe problems washing or dressing | 2 | 0
  Baseline:unable to wash or dress: number analyzed (Participants) | 884 | 439
  Baseline:unable to wash or dress | 4 | 0
  Week 17:no problems washing or dressing: number analyzed (Participants) | 840 | 419
  Week 17:no problems washing or dressing | 752 | 388
  Week 17:slight problems washing or dressing: number analyzed (Participants) | 840 | 419
  Week 17:slight problems washing or dressing | 60 | 26
  Week 17:moderate problems washing or dressing: number analyzed (Participants) | 840 | 419
  Week 17:moderate problems washing or dressing | 21 | 5
  Week 17:severe problems washing or dressing: number analyzed (Participants) | 840 | 419
  Week 17:severe problems washing or dressing | 6 | 0
  Week 17:unable to wash or dress: number analyzed (Participants) | 840 | 419
  Week 17:unable to wash or dress | 1 | 0
  Week 33:no problems washing or dressing: number analyzed (Participants) | 738 | 342
  Week 33:no problems washing or dressing | 642 | 310
  Week 33:slight problems washing or dressing: number analyzed (Participants) | 738 | 342
  Week 33:slight problems washing or dressing | 64 | 20
  Week 33:moderate problems washing or dressing: number analyzed (Participants) | 738 | 342
  Week 33:moderate problems washing or dressing | 21 | 10
  Week 33:severe problems washing or dressing: number analyzed (Participants) | 738 | 342
  Week 33:severe problems washing or dressing | 4 | 1
  Week 33:unable to wash or dress: number analyzed (Participants) | 738 | 342
  Week 33:unable to wash or dress | 7 | 1
  Week 49:no problems washing or dressing: number analyzed (Participants) | 635 | 250
  Week 49:no problems washing or dressing | 546 | 230
  Week 49:slight problems washing or dressing: number analyzed (Participants) | 635 | 250
  Week 49:slight problems washing or dressing | 59 | 9
  Week 49:moderate problems washing or dressing: number analyzed (Participants) | 635 | 250
  Week 49:moderate problems washing or dressing | 23 | 7
  Week 49:severe problems washing or dressing: number analyzed (Participants) | 635 | 250
  Week 49:severe problems washing or dressing | 3 | 3
  Week 49:unable to wash or dress: number analyzed (Participants) | 635 | 250
  Week 49:unable to wash or dress | 4 | 1
  Week 65:no problems washing or dressing: number analyzed (Participants) | 536 | 193
  Week 65:no problems washing or dressing | 453 | 179
  Week 65:slight problems washing or dressing: number analyzed (Participants) | 536 | 193
  Week 65:slight problems washing or dressing | 57 | 11
  Week 65:moderate problems washing or dressing: number analyzed (Participants) | 536 | 193
  Week 65:moderate problems washing or dressing | 14 | 3
  Week 65:severe problems washing or dressing: number analyzed (Participants) | 536 | 193
  Week 65:severe problems washing or dressing | 9 | 0
  Week 65:unable to wash or dress: number analyzed (Participants) | 536 | 193
  Week 65:unable to wash or dress | 3 | 0
  Week 81:no problems washing or dressing: number analyzed (Participants) | 435 | 148
  Week 81:no problems washing or dressing | 356 | 132
  Week 81:slight problems washing or dressing: number analyzed (Participants) | 435 | 148
  Week 81:slight problems washing or dressing | 57 | 11
  Week 81:moderate problems washing or dressing: number analyzed (Participants) | 435 | 148
  Week 81:moderate problems washing or dressing | 17 | 3
  Week 81:severe problems washing or dressing: number analyzed (Participants) | 435 | 148
  Week 81:severe problems washing or dressing | 3 | 1
  Week 81:unable to wash or dress: number analyzed (Participants) | 435 | 148
  Week 81:unable to wash or dress | 2 | 1
  Week 97:no problems washing or dressing: number analyzed (Participants) | 365 | 95
  Week 97:no problems washing or dressing | 292 | 85
  Week 97:slight problems washing or dressing: number analyzed (Participants) | 365 | 95
  Week 97:slight problems washing or dressing | 51 | 8
  Week 97:moderate problems washing or dressing: number analyzed (Participants) | 365 | 95
  Week 97:moderate problems washing or dressing | 16 | 2
  Week 97:severe problems washing or dressing: number analyzed (Participants) | 365 | 95
  Week 97:severe problems washing or dressing | 1 | 0
  Week 97:unable to wash or dress: number analyzed (Participants) | 365 | 95
  Week 97:unable to wash or dress | 5 | 0
  Week 113:no problems washing or dressing: number analyzed (Participants) | 275 | 73
  Week 113:no problems washing or dressing | 214 | 60
  Week 113:slight problems washing or dressing: number analyzed (Participants) | 275 | 73
  Week 113:slight problems washing or dressing | 46 | 7
  Week 113:moderate problems washing or dressing: number analyzed (Participants) | 275 | 73
  Week 113:moderate problems washing or dressing | 11 | 5
  Week 113:severe problems washing or dressing: number analyzed (Participants) | 275 | 73
  Week 113:severe problems washing or dressing | 0 | 0
  Week 113:unable to wash or dress: number analyzed (Participants) | 275 | 73
  Week 113:unable to wash or dress | 4 | 1
  Week 129:no problems washing or dressing: number analyzed (Participants) | 193 | 41
  Week 129:no problems washing or dressing | 147 | 35
  Week 129:slight problems washing or dressing: number analyzed (Participants) | 193 | 41
  Week 129:slight problems washing or dressing | 28 | 5
  Week 129:moderate problems washing or dressing: number analyzed (Participants) | 193 | 41
  Week 129:moderate problems washing or dressing | 16 | 1
  Week 129:severe problems washing or dressing: number analyzed (Participants) | 193 | 41
  Week 129:severe problems washing or dressing | 2 | 0
  Week 129:unable to wash or dress: number analyzed (Participants) | 193 | 41
  Week 129:unable to wash or dress | 0 | 0
  Week 145:no problems washing or dressing: number analyzed (Participants) | 116 | 21
  Week 145:no problems washing or dressing | 92 | 15
  Week 145:slight problems washing or dressing: number analyzed (Participants) | 116 | 21
  Week 145:slight problems washing or dressing | 16 | 5
  Week 145:moderate problems washing or dressing: number analyzed (Participants) | 116 | 21
  Week 145:moderate problems washing or dressing | 6 | 0
  Week 145:severe problems washing or dressing: number analyzed (Participants) | 116 | 21
  Week 145:severe problems washing or dressing | 2 | 0
  Week 145:unable to wash or dress: number analyzed (Participants) | 116 | 21
  Week 145:unable to wash or dress | 0 | 1
  Week 161:no problems washing or dressing: number analyzed (Participants) | 40 | 8
  Week 161:no problems washing or dressing | 33 | 7
  Week 161:slight problems washing or dressing: number analyzed (Participants) | 40 | 8
  Week 161:slight problems washing or dressing | 3 | 0
  Week 161:moderate problems washing or dressing: number analyzed (Participants) | 40 | 8
  Week 161:moderate problems washing or dressing | 2 | 1
  Week 161:severe problems washing or dressing: number analyzed (Participants) | 40 | 8
  Week 161:severe problems washing or dressing | 1 | 0
  Week 161:unable to wash or dress: number analyzed (Participants) | 40 | 8
  Week 161:unable to wash or dress | 1 | 0
  Week 177:no problems washing or dressing: number analyzed (Participants) | 6 | 1
  Week 177:no problems washing or dressing | 3 | 1
  Week 177:slight problems washing or dressing: number analyzed (Participants) | 6 | 1
  Week 177:slight problems washing or dressing | 3 | 0
  Week 177:moderate problems washing or dressing: number analyzed (Participants) | 6 | 1
  Week 177:moderate problems washing or dressing | 0 | 0
  Week 177:severe problems washing or dressing: number analyzed (Participants) | 6 | 1
  Week 177:severe problems washing or dressing | 0 | 0
  Week 171:unable to wash or dress: number analyzed (Participants) | 6 | 1
  Week 171:unable to wash or dress | 0 | 0

13. Secondary Outcome: Number of Participants With European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Usual Activities Domain Score
Description: EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Number of participants with various responses to the usual activities questionnaire are reported.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: The ITT population was defined as all participants randomly assigned to study treatment and was based on randomized treatment assignment regardless of whether or not treatment was administered. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified categories.
Measure: Number; unit: participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
participants
  Baseline:no problems doing usual activities: number analyzed (Participants) | 884 | 439
  Baseline:no problems doing usual activities | 646 | 356
  Baseline:slight problems doing usual activities: number analyzed (Participants) | 884 | 439
  Baseline:slight problems doing usual activities | 167 | 64
  Baseline:moderate problems: number analyzed (Participants) | 884 | 439
  Baseline:moderate problems | 56 | 14
  Baseline:severe problems: number analyzed (Participants) | 884 | 439
  Baseline:severe problems | 10 | 5
  Baseline:unable to do usual activities: number analyzed (Participants) | 884 | 439
  Baseline:unable to do usual activities | 5 | 0
  Week 17:no problems doing usual activities: number analyzed (Participants) | 840 | 419
  Week 17:no problems doing usual activities | 571 | 305
  Week 17:slight problems doing usual activities: number analyzed (Participants) | 840 | 419
  Week 17:slight problems doing usual activities | 181 | 89
  Week 17:moderate problems: number analyzed (Participants) | 840 | 419
  Week 17:moderate problems | 60 | 24
  Week 17:severe problems: number analyzed (Participants) | 840 | 419
  Week 17:severe problems | 21 | 0
  Week 17:unable to do usual activities: number analyzed (Participants) | 840 | 419
  Week 17:unable to do usual activities | 7 | 1
  Week 33:no problems doing usual activities: number analyzed (Participants) | 738 | 342
  Week 33:no problems doing usual activities | 474 | 249
  Week 33:slight problems doing usual activities: number analyzed (Participants) | 738 | 342
  Week 33:slight problems doing usual activities | 170 | 68
  Week 33:moderate problems: number analyzed (Participants) | 738 | 342
  Week 33:moderate problems | 68 | 18
  Week 33:severe problems: number analyzed (Participants) | 738 | 342
  Week 33:severe problems | 21 | 7
  Week 33:unable to do usual activities: number analyzed (Participants) | 738 | 342
  Week 33:unable to do usual activities | 5 | 0
  Week 49:no problems doing usual activities: number analyzed (Participants) | 635 | 250
  Week 49:no problems doing usual activities | 418 | 185
  Week 49:slight problems doing usual activities: number analyzed (Participants) | 635 | 250
  Week 49:slight problems doing usual activities | 137 | 43
  Week 49:moderate problems: number analyzed (Participants) | 635 | 250
  Week 49:moderate problems | 55 | 14
  Week 49:severe problems: number analyzed (Participants) | 635 | 250
  Week 49:severe problems | 20 | 6
  Week 49:unable to do usual activities: number analyzed (Participants) | 635 | 250
  Week 49:unable to do usual activities | 5 | 2
  Week 65:no problems doing usual activities: number analyzed (Participants) | 536 | 193
  Week 65:no problems doing usual activities | 338 | 136
  Week 65:slight problems doing usual activities: number analyzed (Participants) | 536 | 193
  Week 65:slight problems doing usual activities | 123 | 42
  Week 65:moderate problems: number analyzed (Participants) | 536 | 193
  Week 65:moderate problems | 60 | 11
  Week 65:severe problems: number analyzed (Participants) | 536 | 193
  Week 65:severe problems | 5 | 4
  Week 65:unable to do usual activities: number analyzed (Participants) | 536 | 193
  Week 65:unable to do usual activities | 10 | 0
  Week 81:no problems doing usual activities: number analyzed (Participants) | 435 | 148
  Week 81:no problems doing usual activities | 267 | 106
  Week 81:slight problems doing usual activities: number analyzed (Participants) | 435 | 148
  Week 81:slight problems doing usual activities | 105 | 29
  Week 81:moderate problems: number analyzed (Participants) | 435 | 148
  Week 81:moderate problems | 49 | 7
  Week 81:severe problems: number analyzed (Participants) | 435 | 148
  Week 81:severe problems | 10 | 3
  Week 81:unable to do usual activities: number analyzed (Participants) | 435 | 148
  Week 81:unable to do usual activities | 4 | 3
  Week 97:no problems doing usual activities: number analyzed (Participants) | 365 | 95
  Week 97:no problems doing usual activities | 224 | 69
  Week 97:slight problems doing usual activities: number analyzed (Participants) | 365 | 95
  Week 97:slight problems doing usual activities | 90 | 16
  Week 97:moderate problems: number analyzed (Participants) | 365 | 95
  Week 97:moderate problems | 39 | 8
  Week 97:severe problems: number analyzed (Participants) | 365 | 95
  Week 97:severe problems | 9 | 0
  Week 97:unable to do usual activities: number analyzed (Participants) | 365 | 95
  Week 97:unable to do usual activities | 3 | 2
  Week 113:no problems doing usual activities: number analyzed (Participants) | 275 | 73
  Week 113:no problems doing usual activities | 165 | 47
  Week 113:slight problems doing usual activities: number analyzed (Participants) | 275 | 73
  Week 113:slight problems doing usual activities | 69 | 16
  Week 113:moderate problems: number analyzed (Participants) | 275 | 73
  Week 113:moderate problems | 33 | 6
  Week 113:severe problems: number analyzed (Participants) | 275 | 73
  Week 113:severe problems | 5 | 3
  Week 113:unable to do usual activities: number analyzed (Participants) | 275 | 73
  Week 113:unable to do usual activities | 3 | 1
  Week 129: Week :no problems doing usual activities: number analyzed (Participants) | 193 | 41
  Week 129: Week :no problems doing usual activities | 108 | 30
  Week 129 :slight problems doing usual activities: number analyzed (Participants) | 193 | 41
  Week 129 :slight problems doing usual activities | 56 | 8
  Week 129:moderate problems: number analyzed (Participants) | 193 | 41
  Week 129:moderate problems | 26 | 3
  Week 129:severe problems: number analyzed (Participants) | 193 | 41
  Week 129:severe problems | 3 | 0
  Week 129:unable to do usual activities: number analyzed (Participants) | 193 | 41
  Week 129:unable to do usual activities | 0 | 0
  Week 145:no problems doing usual activities: number analyzed (Participants) | 116 | 21
  Week 145:no problems doing usual activities | 67 | 14
  Week 145:slight problems doing usual activities: number analyzed (Participants) | 116 | 21
  Week 145:slight problems doing usual activities | 35 | 4
  Week 145:moderate problems: number analyzed (Participants) | 116 | 21
  Week 145:moderate problems | 11 | 2
  Week 145:severe problems: number analyzed (Participants) | 116 | 21
  Week 145:severe problems | 3 | 1
  Week 145:unable to do usual activities: number analyzed (Participants) | 116 | 21
  Week 145:unable to do usual activities | 0 | 0
  Week 161:no problems doing usual activities: number analyzed (Participants) | 40 | 8
  Week 161:no problems doing usual activities | 23 | 5
  Week 161:slight problems doing usual activities: number analyzed (Participants) | 40 | 8
  Week 161:slight problems doing usual activities | 9 | 2
  Week 161:moderate problems: number analyzed (Participants) | 40 | 8
  Week 161:moderate problems | 5 | 1
  Week 161:severe problems: number analyzed (Participants) | 40 | 8
  Week 161:severe problems | 2 | 0
  Week 161:unable to do usual activities: number analyzed (Participants) | 40 | 8
  Week 161:unable to do usual activities | 1 | 0
  Week 177:no problems doing usual activities: number analyzed (Participants) | 6 | 1
  Week 177:no problems doing usual activities | 3 | 0
  Week 177:slight problems doing usual activities: number analyzed (Participants) | 6 | 1
  Week 177:slight problems doing usual activities | 2 | 1
  Week 177:moderate problems: number analyzed (Participants) | 6 | 1
  Week 177:moderate problems | 1 | 0
  Week 177:severe problems: number analyzed (Participants) | 6 | 1
  Week 177:severe problems | 0 | 0
  Week 177:unable to do usual activities: number analyzed (Participants) | 6 | 1
  Week 177:unable to do usual activities | 0 | 0

14. Secondary Outcome: Number of Participants With European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Pain/Discomfort Domain Score
Description: EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Number of participants with various responses to the pain/discomfort questionnaire are reported.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline:no pain or discomfort: number analyzed (Participants) | 884 | 439
  Baseline:no pain or discomfort | 546 | 292
  Baseline:slight pain or discomfort: number analyzed (Participants) | 884 | 439
  Baseline:slight pain or discomfort | 240 | 117
  Baseline:moderate pain or discomfort: number analyzed (Participants) | 884 | 439
  Baseline:moderate pain or discomfort | 86 | 25
  Baseline:severe pain or discomfort: number analyzed (Participants) | 884 | 439
  Baseline:severe pain or discomfort | 10 | 4
  Baseline:extreme pain or discomfort: number analyzed (Participants) | 884 | 439
  Baseline:extreme pain or discomfort | 2 | 1
  Week 17:no pain or discomfort: number analyzed (Participants) | 840 | 419
  Week 17:no pain or discomfort | 464 | 248
  Week 17:slight pain or discomfort: number analyzed (Participants) | 840 | 419
  Week 17:slight pain or discomfort | 269 | 128
  Week 17: moderate pain or discomfort: number analyzed (Participants) | 840 | 419
  Week 17: moderate pain or discomfort | 92 | 41
  Week 17:severe pain or discomfort: number analyzed (Participants) | 840 | 419
  Week 17:severe pain or discomfort | 13 | 2
  Week 17:extreme pain or discomfort: number analyzed (Participants) | 840 | 419
  Week 17:extreme pain or discomfort | 2 | 0
  Week 33:no pain or discomfort: number analyzed (Participants) | 738 | 342
  Week 33:no pain or discomfort | 405 | 204
  Week 33:slight pain or discomfort: number analyzed (Participants) | 738 | 342
  Week 33:slight pain or discomfort | 237 | 110
  Week 33:moderate pain or discomfort: number analyzed (Participants) | 738 | 342
  Week 33:moderate pain or discomfort | 79 | 21
  Week 33:severe pain or discomfort: number analyzed (Participants) | 738 | 342
  Week 33:severe pain or discomfort | 16 | 7
  Week 33:extreme pain or discomfort: number analyzed (Participants) | 738 | 342
  Week 33:extreme pain or discomfort | 1 | 0
  Week 49:no pain or discomfort: number analyzed (Participants) | 635 | 250
  Week 49:no pain or discomfort | 340 | 134
  Week 49:slight pain or discomfort: number analyzed (Participants) | 635 | 250
  Week 49:slight pain or discomfort | 209 | 82
  Week 49:moderate pain or discomfort: number analyzed (Participants) | 635 | 250
  Week 49:moderate pain or discomfort | 75 | 32
  Week 49:severe pain or discomfort: number analyzed (Participants) | 635 | 250
  Week 49:severe pain or discomfort | 10 | 1
  Week 49:extreme pain or discomfort: number analyzed (Participants) | 635 | 250
  Week 49:extreme pain or discomfort | 1 | 1
  Week 65:no pain or discomfort: number analyzed (Participants) | 536 | 193
  Week 65:no pain or discomfort | 298 | 102
  Week 65:slight pain or discomfort: number analyzed (Participants) | 536 | 193
  Week 65:slight pain or discomfort | 162 | 72
  Week 65:moderate pain or discomfort: number analyzed (Participants) | 536 | 193
  Week 65:moderate pain or discomfort | 61 | 15
  Week 65:severe pain or discomfort: number analyzed (Participants) | 536 | 193
  Week 65:severe pain or discomfort | 11 | 3
  Week 65:extreme pain or discomfort: number analyzed (Participants) | 536 | 193
  Week 65:extreme pain or discomfort | 4 | 1
  Week 81:no pain or discomfort: number analyzed (Participants) | 435 | 148
  Week 81:no pain or discomfort | 231 | 86
  Week 81:slight pain or discomfort: number analyzed (Participants) | 435 | 148
  Week 81:slight pain or discomfort | 133 | 45
  Week 81:moderate pain or discomfort: number analyzed (Participants) | 435 | 148
  Week 81:moderate pain or discomfort | 61 | 13
  Week 81 :severe pain or discomfort: number analyzed (Participants) | 435 | 148
  Week 81 :severe pain or discomfort | 10 | 2
  Week 81:extreme pain or discomfort: number analyzed (Participants) | 435 | 148
  Week 81:extreme pain or discomfort | 0 | 2
  Week 97:no pain or discomfort: number analyzed (Participants) | 365 | 95
  Week 97:no pain or discomfort | 202 | 58
  Week 97:slight pain or discomfort: number analyzed (Participants) | 365 | 95
  Week 97:slight pain or discomfort | 115 | 28
  Week 97:moderate pain or discomfort: number analyzed (Participants) | 365 | 95
  Week 97:moderate pain or discomfort | 43 | 7
  Week 97:severe pain or discomfort: number analyzed (Participants) | 365 | 95
  Week 97:severe pain or discomfort | 5 | 2
  Week 97:extreme pain or discomfort: number analyzed (Participants) | 365 | 95
  Week 97:extreme pain or discomfort | 0 | 0
  Week 113:no pain or discomfort: number analyzed (Participants) | 275 | 73
  Week 113:no pain or discomfort | 152 | 47
  Week 113:slight pain or discomfort: number analyzed (Participants) | 275 | 73
  Week 113:slight pain or discomfort | 80 | 19
  Week 113:moderate pain or discomfort: number analyzed (Participants) | 275 | 73
  Week 113:moderate pain or discomfort | 37 | 5
  Week 113:severe pain or discomfort: number analyzed (Participants) | 275 | 73
  Week 113:severe pain or discomfort | 6 | 2
  Week 113:extreme pain or discomfort: number analyzed (Participants) | 275 | 73
  Week 113:extreme pain or discomfort | 0 | 0
  Week 129:no pain or discomfort: number analyzed (Participants) | 193 | 41
  Week 129:no pain or discomfort | 108 | 27
  Week 129:slight pain or discomfort: number analyzed (Participants) | 193 | 41
  Week 129:slight pain or discomfort | 55 | 11
  Week 129:moderate pain or discomfort: number analyzed (Participants) | 193 | 41
  Week 129:moderate pain or discomfort | 28 | 3
  Week 129:severe pain or discomfort: number analyzed (Participants) | 193 | 41
  Week 129:severe pain or discomfort | 2 | 0
  Week 129:extreme pain or discomfort: number analyzed (Participants) | 193 | 41
  Week 129:extreme pain or discomfort | 0 | 0
  Week 145:no pain or discomfort: number analyzed (Participants) | 116 | 21
  Week 145:no pain or discomfort | 62 | 12
  Week 145:slight pain or discomfort: number analyzed (Participants) | 116 | 21
  Week 145:slight pain or discomfort | 38 | 8
  Week 145:moderate pain or discomfort: number analyzed (Participants) | 116 | 21
  Week 145:moderate pain or discomfort | 15 | 1
  Week 145:severe pain or discomfort: number analyzed (Participants) | 116 | 21
  Week 145:severe pain or discomfort | 1 | 0
  Week 145:extreme pain or discomfort: number analyzed (Participants) | 116 | 21
  Week 145:extreme pain or discomfort | 0 | 0
  Week 161:no pain or discomfort: number analyzed (Participants) | 40 | 8
  Week 161:no pain or discomfort | 24 | 2
  Week 161:slight pain or discomfort: number analyzed (Participants) | 40 | 8
  Week 161:slight pain or discomfort | 8 | 5
  Week 161:moderate pain or discomfort: number analyzed (Participants) | 40 | 8
  Week 161:moderate pain or discomfort | 5 | 1
  Week 161:severe pain or discomfort: number analyzed (Participants) | 40 | 8
  Week 161:severe pain or discomfort | 3 | 0
  Week 161:extreme pain or discomfort: number analyzed (Participants) | 40 | 8
  Week 161:extreme pain or discomfort | 0 | 0
  Week 177:no pain or discomfort: number analyzed (Participants) | 6 | 1
  Week 177:no pain or discomfort | 3 | 0
  Week 177:slight pain or discomfort: number analyzed (Participants) | 6 | 1
  Week 177:slight pain or discomfort | 1 | 1
  Week 177:moderate pain or discomfort: number analyzed (Participants) | 6 | 1
  Week 177:moderate pain or discomfort | 2 | 0
  Week 177:severe pain or discomfort: number analyzed (Participants) | 6 | 1
  Week 177:severe pain or discomfort | 0 | 0
  Week 177:extreme pain or discomfort: number analyzed (Participants) | 6 | 1
  Week 177:extreme pain or discomfort | 0 | 0

15. Secondary Outcome: Number of Participants With European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Anxiety/ Depression Domain Score
Description: EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. Number of participants with various responses to the anxiety/depression questionnaire are reported.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline:not anxious or depressed: number analyzed (Participants) | 884 | 439
  Baseline:not anxious or depressed | 595 | 310
  Baseline:slightly anxious or depressed: number analyzed (Participants) | 884 | 439
  Baseline:slightly anxious or depressed | 231 | 100
  Baseline:moderately anxious or depressed: number analyzed (Participants) | 884 | 439
  Baseline:moderately anxious or depressed | 51 | 24
  Baseline:severely anxious or depressed: number analyzed (Participants) | 884 | 439
  Baseline:severely anxious or depressed | 6 | 5
  Baseline:extremely anxious or depressed: number analyzed (Participants) | 884 | 439
  Baseline:extremely anxious or depressed | 1 | 0
  Week 17:not anxious or depressed: number analyzed (Participants) | 840 | 419
  Week 17:not anxious or depressed | 517 | 265
  Week 17:slightly anxious or depressed: number analyzed (Participants) | 840 | 419
  Week 17:slightly anxious or depressed | 251 | 119
  Week 17:moderately anxious or depressed: number analyzed (Participants) | 840 | 419
  Week 17:moderately anxious or depressed | 62 | 31
  Week 17:severely anxious or depressed: number analyzed (Participants) | 840 | 419
  Week 17:severely anxious or depressed | 7 | 4
  Week 17:extremely anxious or depressed: number analyzed (Participants) | 840 | 419
  Week 17:extremely anxious or depressed | 3 | 0
  Week 33:not anxious or depressed: number analyzed (Participants) | 738 | 342
  Week 33:not anxious or depressed | 458 | 223
  Week 33:slightly anxious or depressed: number analyzed (Participants) | 738 | 342
  Week 33:slightly anxious or depressed | 208 | 89
  Week 33:moderately anxious or depressed: number analyzed (Participants) | 738 | 342
  Week 33:moderately anxious or depressed | 61 | 23
  Week 33:severely anxious or depressed: number analyzed (Participants) | 738 | 342
  Week 33:severely anxious or depressed | 9 | 5
  Week 33:extremely anxious or depressed: number analyzed (Participants) | 738 | 342
  Week 33:extremely anxious or depressed | 2 | 2
  Week 49:not anxious or depressed: number analyzed (Participants) | 635 | 250
  Week 49:not anxious or depressed | 410 | 155
  Week 49:slightly anxious or depressed: number analyzed (Participants) | 635 | 250
  Week 49:slightly anxious or depressed | 172 | 72
  Week 49:moderately anxious or depressed: number analyzed (Participants) | 635 | 250
  Week 49:moderately anxious or depressed | 41 | 20
  Week 49:severely anxious or depressed: number analyzed (Participants) | 635 | 250
  Week 49:severely anxious or depressed | 8 | 2
  Week 49:extremely anxious or depressed: number analyzed (Participants) | 635 | 250
  Week 49:extremely anxious or depressed | 4 | 1
  Week 65:not anxious or depressed: number analyzed (Participants) | 536 | 193
  Week 65:not anxious or depressed | 336 | 128
  Week 65:slightly anxious or depressed: number analyzed (Participants) | 536 | 193
  Week 65:slightly anxious or depressed | 149 | 56
  Week 65:moderately anxious or depressed: number analyzed (Participants) | 536 | 193
  Week 65:moderately anxious or depressed | 43 | 8
  Week 65:severely anxious or depressed: number analyzed (Participants) | 536 | 193
  Week 65:severely anxious or depressed | 8 | 1
  Week 65:extremely anxious or depressed: number analyzed (Participants) | 536 | 193
  Week 65:extremely anxious or depressed | 0 | 0
  Week 81:not anxious or depressed: number analyzed (Participants) | 435 | 148
  Week 81:not anxious or depressed | 288 | 86
  Week 81:slightly anxious or depressed: number analyzed (Participants) | 435 | 148
  Week 81:slightly anxious or depressed | 106 | 48
  Week 81:moderately anxious or depressed: number analyzed (Participants) | 435 | 148
  Week 81:moderately anxious or depressed | 34 | 9
  Week 81:severely anxious or depressed: number analyzed (Participants) | 435 | 148
  Week 81:severely anxious or depressed | 7 | 3
  Week 81:extremely anxious or depressed: number analyzed (Participants) | 435 | 148
  Week 81:extremely anxious or depressed | 0 | 2
  Week 97:not anxious or depressed: number analyzed (Participants) | 365 | 95
  Week 97:not anxious or depressed | 220 | 61
  Week 97:slightly anxious or depressed: number analyzed (Participants) | 365 | 95
  Week 97:slightly anxious or depressed | 114 | 27
  Week 97:moderately anxious or depressed: number analyzed (Participants) | 365 | 95
  Week 97:moderately anxious or depressed | 26 | 6
  Week 97:severely anxious or depressed: number analyzed (Participants) | 365 | 95
  Week 97:severely anxious or depressed | 4 | 0
  Week 97:extremely anxious or depressed: number analyzed (Participants) | 365 | 95
  Week 97:extremely anxious or depressed | 1 | 1
  Week 113:not anxious or depressed: number analyzed (Participants) | 275 | 73
  Week 113:not anxious or depressed | 167 | 43
  Week 113:slightly anxious or depressed: number analyzed (Participants) | 275 | 73
  Week 113:slightly anxious or depressed | 87 | 27
  Week 113:moderately anxious or depressed: number analyzed (Participants) | 275 | 73
  Week 113:moderately anxious or depressed | 18 | 3
  Week 113:severely anxious or depressed: number analyzed (Participants) | 275 | 73
  Week 113:severely anxious or depressed | 3 | 0
  Week 113:extremely anxious or depressed: number analyzed (Participants) | 275 | 73
  Week 113:extremely anxious or depressed | 0 | 0
  Week 129:not anxious or depressed: number analyzed (Participants) | 193 | 41
  Week 129:not anxious or depressed | 121 | 28
  Week 129:slightly anxious or depressed: number analyzed (Participants) | 193 | 41
  Week 129:slightly anxious or depressed | 51 | 10
  Week 129:moderately anxious or depressed: number analyzed (Participants) | 193 | 41
  Week 129:moderately anxious or depressed | 18 | 2
  Week 129:severely anxious or depressed: number analyzed (Participants) | 193 | 41
  Week 129:severely anxious or depressed | 2 | 1
  Week 129:extremely anxious or depressed: number analyzed (Participants) | 193 | 41
  Week 129:extremely anxious or depressed | 1 | 0
  Week 145:not anxious or depressed: number analyzed (Participants) | 116 | 21
  Week 145:not anxious or depressed | 73 | 12
  Week 145:slightly anxious or depressed: number analyzed (Participants) | 116 | 21
  Week 145:slightly anxious or depressed | 30 | 8
  Week 145:moderately anxious or depressed: number analyzed (Participants) | 116 | 21
  Week 145:moderately anxious or depressed | 10 | 1
  Week 145:severely anxious or depressed: number analyzed (Participants) | 116 | 21
  Week 145:severely anxious or depressed | 2 | 0
  Week 145:extremely anxious or depressed: number analyzed (Participants) | 116 | 21
  Week 145:extremely anxious or depressed | 1 | 0
  Week 161:not anxious or depressed: number analyzed (Participants) | 40 | 8
  Week 161:not anxious or depressed | 23 | 3
  Week 161:slightly anxious or depressed: number analyzed (Participants) | 40 | 8
  Week 161:slightly anxious or depressed | 16 | 4
  Week 161:moderately anxious or depressed: number analyzed (Participants) | 40 | 8
  Week 161:moderately anxious or depressed | 0 | 1
  Week 161:severely anxious or depressed: number analyzed (Participants) | 40 | 8
  Week 161:severely anxious or depressed | 0 | 0
  Week 161:extremely anxious or depressed: number analyzed (Participants) | 40 | 8
  Week 161:extremely anxious or depressed | 1 | 0
  Week 177:not anxious or depressed: number analyzed (Participants) | 933 | 1
  Week 177:not anxious or depressed | 2 | 1
  Week 177:slightly anxious or depressed: number analyzed (Participants) | 6 | 1
  Week 177:slightly anxious or depressed | 2 | 0
  Week 177:moderately anxious or depressed: number analyzed (Participants) | 6 | 1
  Week 177:moderately anxious or depressed | 2 | 0
  Week 177:severely anxious or depressed: number analyzed (Participants) | 6 | 1
  Week 177:severely anxious or depressed | 0 | 0
  Week 177:extremely anxious or depressed: number analyzed (Participants) | 6 | 1
  Week 177:extremely anxious or depressed | 0 | 0

16. Secondary Outcome: European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Overall Health Status Visual Analog Score (VAS)
Description: EQ-5D-5L is a standardized instrument that measures health-related quality of life for men with prostate cancer. EQ-5D consists of EQ-5D descriptive system and EQ VAS. EQ-5D-5L-VAS records participant's self-rated health on a vertical VAS that allows them to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable), higher scores indicating a better health state.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
units on a scale
  Baseline: number analyzed (Participants) | 884 | 439
  Baseline | 76.2 (16.92) | 77.5 (15.97)
  Week 17: number analyzed (Participants) | 840 | 419
  Week 17 | 74.7 (17.19) | 74.9 (16.79)
  Week 33: number analyzed (Participants) | 738 | 342
  Week 33 | 74.6 (16.69) | 74.0 (17.51)
  Week 49: number analyzed (Participants) | 635 | 250
  Week 49 | 74.7 (18.02) | 73.7 (18.28)
  Week 65: number analyzed (Participants) | 536 | 193
  Week 65 | 74.5 (17.79) | 73.0 (17.11)
  Week 81: number analyzed (Participants) | 435 | 148
  Week 81 | 75.5 (17.06) | 73.3 (16.82)
  Week 97: number analyzed (Participants) | 365 | 95
  Week 97 | 74.4 (17.39) | 75.2 (17.88)
  Week 113: number analyzed (Participants) | 275 | 73
  Week 113 | 73.6 (18.05) | 74.7 (15.06)
  Week 129: number analyzed (Participants) | 193 | 41
  Week 129 | 72.8 (18.25) | 77.1 (12.83)
  Week 145: number analyzed (Participants) | 116 | 21
  Week 145 | 75.3 (17.02) | 74.2 (18.13)
  Week 161: number analyzed (Participants) | 40 | 8
  Week 161 | 74.6 (21.28) | 73.8 (17.60)
  Week 177: number analyzed (Participants) | 6 | 1
  Week 177 | 74.5 (19.31) | 69.0

17. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 31
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 31 are reported. Question 31 was following: "Have you had to urinate frequently during the day?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 285 | 162
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 348 | 160
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 207 | 92
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 44 | 25
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 275 | 134
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 324 | 168
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 194 | 90
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 46 | 27
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 236 | 105
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 285 | 145
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 176 | 70
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 40 | 21
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 200 | 82
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 260 | 92
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 148 | 67
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 27 | 9
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 172 | 54
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 209 | 79
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 125 | 48
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 30 | 12
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 141 | 46
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 181 | 60
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 92 | 31
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 20 | 11
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 118 | 33
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 146 | 40
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 80 | 19
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 21 | 3
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 101 | 17
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 112 | 40
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 46 | 14
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 16 | 2
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 70 | 11
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 79 | 16
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 39 | 10
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 4 | 4
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 42 | 2
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 51 | 14
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 20 | 4
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 3 | 1
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 9 | 2
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 20 | 4
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 7 | 1
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 4 | 1
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 0 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 4 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 2 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

18. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 32
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 32 are reported. Question 32 was following: "Have you had to urinate frequently at night?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 193 | 108
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 423 | 195
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 200 | 103
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 68 | 33
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 194 | 88
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 407 | 199
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 184 | 98
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 54 | 34
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 173 | 83
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 351 | 161
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 169 | 69
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 44 | 28
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 148 | 59
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 313 | 116
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 141 | 59
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 33 | 16
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 118 | 41
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 266 | 89
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 111 | 48
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 41 | 15
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 91 | 38
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 231 | 60
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 89 | 38
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 23 | 12
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 88 | 19
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 169 | 53
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 82 | 19
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 26 | 4
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 67 | 16
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 137 | 32
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 54 | 23
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 17 | 2
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 50 | 9
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 97 | 18
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 37 | 10
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 8 | 4
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 31 | 2
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 59 | 14
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 24 | 5
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 2 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 9 | 0
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 23 | 7
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 5 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 3 | 1
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 2 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 2 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 2 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

19. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 33
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 33 are reported. Question 33 was following: "When you felt the urge to pass urine, did you have to hurry to get to the toilet?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 406 | 197
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 266 | 147
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 150 | 70
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 62 | 25
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 350 | 191
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 297 | 150
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 127 | 55
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 65 | 23
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 279 | 147
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 278 | 126
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 126 | 48
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 54 | 20
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 272 | 100
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 222 | 95
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 96 | 38
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 45 | 17
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 213 | 76
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 213 | 72
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 71 | 31
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 39 | 14
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 181 | 63
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 157 | 52
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 69 | 27
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 27 | 6
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 146 | 40
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 131 | 40
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 59 | 12
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 29 | 3
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 114 | 29
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 106 | 34
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 40 | 9
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 15 | 1
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 86 | 10
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 72 | 21
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 26 | 6
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 8 | 4
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 51 | 5
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 39 | 12
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 21 | 4
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 5 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 17 | 0
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 19 | 5
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 3 | 3
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 1 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 2 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 1 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 3 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

20. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 34
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 34 are reported. Question 34 was following: "Was it difficult for you to get enough sleep, because you needed to get up frequently at night to urinate?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 479 | 235
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 273 | 146
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 93 | 40
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 39 | 18
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 437 | 214
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 295 | 144
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 75 | 45
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 32 | 16
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 392 | 180
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 246 | 112
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 75 | 33
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 24 | 16
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 340 | 119
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 211 | 94
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 65 | 28
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 19 | 9
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 286 | 92
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 183 | 67
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 47 | 29
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 20 | 5
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 221 | 70
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 165 | 55
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 37 | 18
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 11 | 5
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 185 | 47
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 122 | 33
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 43 | 14
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 15 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 135 | 31
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 102 | 33
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 29 | 7
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 9 | 2
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 103 | 13
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 67 | 23
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 19 | 4
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 3 | 1
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 59 | 9
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 44 | 10
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 11 | 1
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 2 | 1
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 21 | 2
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 16 | 5
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 3 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 1
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 3 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 1 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 2 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

21. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 35
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 35 are reported. Question 35 was following: "Have you had difficulty going out of the house because you needed to be close to a toilet?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 646 | 330
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 177 | 84
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 45 | 18
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 16 | 7
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 604 | 295
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 174 | 100
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 46 | 15
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 15 | 9
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 501 | 242
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 171 | 74
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 50 | 20
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 15 | 5
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 436 | 174
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 153 | 53
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 38 | 20
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 8 | 3
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 369 | 132
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 125 | 50
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 28 | 9
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 14 | 2
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 308 | 105
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 94 | 35
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 23 | 8
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 9 | 0
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 241 | 67
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 91 | 21
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 26 | 6
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 7 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 180 | 47
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 70 | 21
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 18 | 5
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 7 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 131 | 26
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 48 | 13
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 8 | 1
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 5 | 1
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 74 | 13
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 36 | 6
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 6 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 2
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 24 | 4
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 13 | 4
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 3 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 3 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 3 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

22. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 36
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 36 are reported. Question 36 was following: "Have you had any unintentional release (leakage) of urine?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 550 | 283
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 273 | 124
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 36 | 20
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 25 | 12
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 511 | 255
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 264 | 126
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 39 | 27
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 25 | 11
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 428 | 208
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 246 | 104
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 34 | 19
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 29 | 10
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 369 | 146
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 209 | 78
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 41 | 22
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 16 | 4
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 307 | 115
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 170 | 66
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 47 | 8
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 12 | 4
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 248 | 93
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 158 | 41
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 23 | 11
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 5 | 3
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 195 | 55
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 134 | 33
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 25 | 7
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 11 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 160 | 42
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 91 | 28
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 17 | 3
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 7 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 109 | 22
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 68 | 13
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 13 | 5
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 2 | 1
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 58 | 9
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 45 | 11
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 10 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 3 | 1
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 18 | 3
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 21 | 4
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 0 | 1
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 1 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 1 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 3 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 1 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 1 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

23. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 37
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 37 are reported. Question 37 was following: "Did you have pain when you urinated?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 775 | 380
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 92 | 47
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 10 | 8
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 7 | 4
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 762 | 351
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 65 | 58
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 12 | 8
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 0 | 2
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 662 | 291
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 63 | 39
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 11 | 8
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 1 | 3
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 577 | 209
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 49 | 34
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 6 | 3
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 3 | 4
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 492 | 161
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 32 | 29
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 9 | 2
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 3 | 1
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 389 | 119
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 40 | 27
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 4 | 2
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 1 | 0
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 332 | 84
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 28 | 11
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 4 | 0
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 1 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 247 | 57
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 26 | 13
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 1 | 3
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 1 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 173 | 34
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 16 | 7
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 1 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 2 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 102 | 15
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 14 | 6
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 0 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 36 | 6
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 3 | 1
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 1
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 6 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

24. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 38
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 38 are reported. Question 38 was following: "Has wearing an incontinence aid been a problem for you?". This question was answered by only those participants who wore incontinence aid.
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 144 | 67
  Baseline: not at all | 83 | 37
  Baseline: a little: number analyzed (Participants) | 144 | 67
  Baseline: a little | 40 | 19
  Baseline: quite a bit: number analyzed (Participants) | 144 | 67
  Baseline: quite a bit | 15 | 3
  Baseline: very much: number analyzed (Participants) | 144 | 67
  Baseline: very much | 6 | 8
  Baseline: not answered: number analyzed (Participants) | 144 | 67
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 77 | 34
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 48 | 21
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 15 | 7
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 6 | 6
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 693 | 351
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 76 | 30
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 47 | 28
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 16 | 4
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 5 | 4
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 593 | 275
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 73 | 18
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 43 | 16
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 12 | 9
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 4 | 2
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 503 | 205
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 63 | 12
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 40 | 17
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 9 | 5
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 3 | 1
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 421 | 158
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 52 | 15
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 33 | 9
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 10 | 1
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 3 | 3
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 336 | 120
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 50 | 8
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 28 | 8
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 7 | 2
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 3 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 277 | 77
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 31 | 12
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 18 | 7
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 8 | 2
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 2 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 216 | 52
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 27 | 5
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 18 | 5
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 2 | 1
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 0 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 145 | 30
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 16 | 2
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 10 | 4
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 5 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 85 | 15
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 10 | 1
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 3 | 2
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 1
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 26 | 4
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 3 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 1 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 2 | 1

25. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 39
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 39 are reported. Question 39 was following: "Have your daily activities been limited by your urinary problems?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 666 | 338
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 173 | 80
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 35 | 11
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 10 | 10
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 632 | 305
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 160 | 99
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 36 | 6
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 11 | 9
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 523 | 242
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 172 | 79
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 31 | 14
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 11 | 6
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 444 | 173
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 152 | 58
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 31 | 18
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 8 | 1
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 382 | 128
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 124 | 51
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 20 | 12
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 10 | 2
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 310 | 103
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 98 | 35
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 21 | 8
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 5 | 2
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 242 | 72
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 100 | 18
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 18 | 4
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 5 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 188 | 54
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 71 | 14
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 13 | 3
  Week 113: very much: number analyzed (Participants) | 275 | 93
  Week 113: very much | 3 | 2
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 127 | 25
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 55 | 14
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 7 | 1
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 3 | 1
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 77 | 11
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 34 | 9
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 4 | 1
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 1 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 27 | 2
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 10 | 6
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 3 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 3 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 3 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

26. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 40
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 40 are reported. Question 40 was following: "Have your daily activities been limited by your bowel problems?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 758 | 393
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 112 | 40
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 9 | 4
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 5 | 2
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 707 | 352
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 107 | 57
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 19 | 6
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 6 | 4
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 621 | 292
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 98 | 40
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 14 | 8
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 4 | 1
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 525 | 211
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 88 | 29
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 20 | 7
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 2 | 3
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 441 | 165
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 78 | 24
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 11 | 3
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 6 | 1
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 360 | 121
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 56 | 23
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 17 | 3
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 1 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 289 | 84
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 58 | 11
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 17 | 0
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 1 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 219 | 62
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 46 | 11
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 8 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 2 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 153 | 36
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 33 | 5
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 5 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 1 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 93 | 17
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 19 | 4
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 4 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 29 | 8
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 9 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 2 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 4 | 1
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 2 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

27. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 41
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 41 are reported. Question 41 was following: "Have you had any unintentional release (leakage) of stools?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 794 | 404
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 78 | 32
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 11 | 2
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 1 | 1
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 751 | 372
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 79 | 43
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 8 | 3
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 1 | 1
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 638 | 307
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 92 | 32
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 4 | 1
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 3 | 1
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 554 | 221
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 73 | 25
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 5 | 4
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 3 | 0
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 467 | 175
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 57 | 16
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 9 | 1
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 3 | 1
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 380 | 136
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 51 | 12
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 2 | 0
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 1 | 0
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 315 | 86
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 47 | 9
  Week 97: quite a bit: number analyzed (Participants) | 933 | 95
  Week 97: quite a bit | 3 | 0
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 0 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 233 | 66
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 40 | 7
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 2 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 0 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 167 | 39
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 25 | 2
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 0 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 0 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 93 | 20
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 22 | 1
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 0 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 1 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 30 | 8
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 9 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 0 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 1 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 4 | 1
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 2 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

28. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 42
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 42 are reported. Question 42 was following: "Have you had blood in your stools?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 836 | 422
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 48 | 17
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 0 | 0
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 0 | 0
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 801 | 399
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 36 | 18
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 2 | 2
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 0 | 0
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 707 | 330
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 29 | 11
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 1 | 0
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 0 | 0
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 608 | 245
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 27 | 5
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 0 | 0
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 0 | 0
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 514 | 180
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 19 | 13
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 3 | 0
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 0 | 0
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 420 | 143
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 14 | 4
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 0 | 1
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 0 | 0
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 357 | 93
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 8 | 2
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 0 | 0
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 0 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 262 | 72
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 13 | 1
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 0 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 0 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 186 | 41
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 5 | 0
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 1 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 0 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 114 | 21
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 2 | 0
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 0 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 38 | 8
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 2 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 0 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 6 | 1
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

29. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 43
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 43 are reported. Question 43 was following: "Did you have a bloated feeling in your abdomen?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 667 | 320
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 190 | 103
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 22 | 16
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 5 | 0
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 601 | 283
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 199 | 121
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 31 | 13
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 8 | 2
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 526 | 235
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 183 | 95
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 22 | 8
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 6 | 3
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 449 | 174
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 163 | 63
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 20 | 11
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 3 | 2
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 381 | 135
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 132 | 51
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 19 | 7
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 4 | 0
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 304 | 103
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 110 | 44
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 18 | 1
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 2 | 0
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 258 | 72
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 87 | 23
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 19 | 0
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 1 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 199 | 55
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 66 | 18
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 9 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 1 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 139 | 25
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 43 | 16
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 8 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 2 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 87 | 13
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 24 | 8
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 4 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 1 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 33 | 6
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 7 | 2
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 0 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 4 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 2 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

30. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 44
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 44 are reported. Question 44 was following: "Did you have hot flushes?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 374 | 177
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 314 | 166
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 151 | 68
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 45 | 28
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 265 | 182
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 311 | 153
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 189 | 62
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 74 | 22
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 253 | 144
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 268 | 116
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 155 | 60
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 61 | 21
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 227 | 112
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 235 | 94
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 130 | 30
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 43 | 14
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 203 | 79
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 194 | 77
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 104 | 30
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 35 | 7
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 175 | 69
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 157 | 58
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 75 | 16
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 27 | 5
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 155 | 48
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 126 | 34
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 57 | 12
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 27 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 114 | 33
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 102 | 24
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 44 | 14
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 15 | 2
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 84 | 22
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 74 | 16
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 23 | 3
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 11 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 45 | 10
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 46 | 10
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 18 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 7 | 1
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 18 | 3
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 14 | 3
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 5 | 2
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 3 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 3 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 1 | 1
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 2 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

31. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 45
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 45 are reported. Question 45 was following: "Have you had sore or enlarged nipples or breasts?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 688 | 333
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 146 | 80
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 38 | 24
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 12 | 2
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 626 | 315
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 160 | 80
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 39 | 18
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 14 | 6
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 526 | 260
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 164 | 62
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 34 | 15
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 13 | 4
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 444 | 188
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 138 | 52
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 41 | 5
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 12 | 5
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 371 | 149
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 119 | 37
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 31 | 7
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 15 | 0
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 306 | 115
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 84 | 26
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 34 | 6
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 10 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 239 | 80
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 92 | 13
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 30 | 1
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 4 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 190 | 55
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 62 | 12
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 19 | 5
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 4 | 1
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 128 | 30
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 51 | 8
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 9 | 3
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 4 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 78 | 17
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 29 | 3
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 7 | 1
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 2 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 26 | 4
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 11 | 3
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 2 | 1
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 2 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 2 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 2 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

32. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 46
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 46 are reported. Question 46 was following: "Have you had swelling in your legs or ankles?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 663 | 323
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 189 | 89
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 22 | 22
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 10 | 5
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 625 | 284
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 179 | 112
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 30 | 21
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 5 | 2
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 530 | 243
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 159 | 76
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 41 | 20
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 7 | 2
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 453 | 176
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 155 | 58
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 23 | 15
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 4 | 1
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 378 | 135
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 127 | 48
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 27 | 10
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 4 | 0
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 301 | 104
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 102 | 36
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 27 | 7
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 4 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 259 | 69
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 79 | 20
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 19 | 5
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 8 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 191 | 40
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 65 | 27
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 16 | 6
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 3 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 134 | 27
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 48 | 14
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 8 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 2 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 76 | 15
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 34 | 5
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 5 | 1
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 1 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 31 | 6
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 8 | 2
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 3 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 3 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 1
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

33. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 47
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 47 are reported. Question 47 was following: "Has weight loss been a problem for you?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 820 | 399
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 48 | 25
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 10 | 10
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 6 | 5
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 733 | 375
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 81 | 28
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 15 | 13
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 10 | 3
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 643 | 296
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 72 | 35
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 13 | 5
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 9 | 5
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 553 | 215
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 61 | 29
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 15 | 3
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 6 | 3
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 479 | 168
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 39 | 20
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 11 | 4
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 7 | 1
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 371 | 136
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 46 | 10
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 14 | 1
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 3 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 314 | 84
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 36 | 10
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 10 | 0
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 5 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 235 | 62
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 27 | 8
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 9 | 1
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 4 | 2
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 169 | 37
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 17 | 4
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 5 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 1 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 95 | 20
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 17 | 1
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 4 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 34 | 8
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 5 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 5 | 1
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 1 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

34. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 48
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 48 are reported. Question 48 was following: "Has weight gain been a problem for you?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 677 | 315
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 153 | 95
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 40 | 16
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 14 | 13
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 674 | 316
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 118 | 74
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 30 | 19
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 17 | 10
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 570 | 259
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 133 | 59
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 21 | 18
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 13 | 5
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 479 | 193
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 125 | 44
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 18 | 10
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 13 | 3
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 410 | 155
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 92 | 27
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 26 | 9
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 8 | 2
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 327 | 115
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 71 | 27
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 28 | 5
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 8 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 267 | 76
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 70 | 16
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 24 | 2
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 4 | 1
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 200 | 60
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 56 | 10
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 10 | 3
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 9 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 156 | 32
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 27 | 8
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 5 | 1
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 4 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 89 | 16
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 18 | 5
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 7 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 2 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 31 | 6
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 6 | 2
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 2 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 2 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 3 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 1 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

35. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 49
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 49 are reported. Question 49 was following: "Have you felt less masculine as a result of your illness or treatment?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 435 | 214
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 234 | 131
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 138 | 59
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 77 | 35
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 400 | 210
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 244 | 115
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 109 | 57
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 86 | 37
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 345 | 167
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 207 | 107
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 109 | 38
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 76 | 29
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 302 | 127
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 187 | 68
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 84 | 36
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 62 | 19
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 263 | 90
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 142 | 57
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 71 | 24
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 60 | 22
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 206 | 74
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 124 | 38
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 57 | 17
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 47 | 19
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 175 | 46
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 98 | 28
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 47 | 10
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 45 | 11
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 136 | 31
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 78 | 27
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 30 | 8
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 31 | 7
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 91 | 18
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 49 | 16
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 27 | 5
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 25 | 2
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 59 | 9
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 31 | 9
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 18 | 1
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 8 | 2
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 18 | 2
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 15 | 3
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 3 | 1
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 4 | 2
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 3 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 3 | 1
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

36. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 50
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 50 are reported. Question 50 was following: "To what extent were you interested in sex?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 586 | 291
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 204 | 101
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 67 | 32
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 27 | 15
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 637 | 293
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 136 | 92
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 45 | 20
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 21 | 14
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 542 | 251
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 136 | 66
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 37 | 18
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 22 | 6
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 483 | 180
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 106 | 50
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 33 | 12
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 13 | 8
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 417 | 143
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 78 | 37
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 27 | 9
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 14 | 4
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 320 | 114
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 76 | 24
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 26 | 9
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 12 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 286 | 65
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 52 | 19
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 20 | 8
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 7 | 3
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 218 | 59
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 36 | 11
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 14 | 1
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 7 | 2
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 156 | 33
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 24 | 6
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 9 | 2
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 3 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 92 | 14
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 16 | 3
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 7 | 4
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 1 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 30 | 5
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 5 | 2
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 4 | 1
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 1 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 4 | 1
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 1 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 1 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

37. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 51
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 51 are reported. Question 51 was following: "To what extent were you sexually active (with or without intercourse)?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 884 | 439
  Baseline: not at all | 735 | 374
  Baseline: a little: number analyzed (Participants) | 884 | 439
  Baseline: a little | 98 | 38
  Baseline: quite a bit: number analyzed (Participants) | 884 | 439
  Baseline: quite a bit | 41 | 19
  Baseline: very much: number analyzed (Participants) | 884 | 439
  Baseline: very much | 10 | 8
  Baseline: not answered: number analyzed (Participants) | 884 | 439
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 734 | 354
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 71 | 44
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 24 | 13
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 10 | 8
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 0 | 0
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 642 | 299
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 68 | 28
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 20 | 9
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 7 | 5
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 0 | 0
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 569 | 214
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 46 | 26
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 15 | 6
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 5 | 4
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 0 | 0
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 485 | 170
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 37 | 14
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 12 | 7
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 2 | 2
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 0 | 0
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 381 | 130
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 32 | 13
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 15 | 5
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 6 | 0
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 0 | 0
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 333 | 79
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 20 | 12
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 9 | 4
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 3 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 0 | 0
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 250 | 68
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 16 | 3
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 6 | 2
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 3 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 0 | 0
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 176 | 37
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 8 | 3
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 5 | 1
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 3 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 0 | 0
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 106 | 17
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 4 | 3
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 5 | 1
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 1 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 0 | 0
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 35 | 6
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 3 | 2
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 1 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 0 | 0
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 5 | 1
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 1 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 0 | 0

38. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 52
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 52 are reported. Question 52 was following: "To what extent was sex enjoyable for you?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 50 | 24
  Baseline: not at all | 5 | 6
  Baseline: a little: number analyzed (Participants) | 50 | 24
  Baseline: a little | 23 | 11
  Baseline: quite a bit: number analyzed (Participants) | 50 | 24
  Baseline: quite a bit | 14 | 5
  Baseline: very much: number analyzed (Participants) | 50 | 24
  Baseline: very much | 8 | 2
  Baseline: not answered: number analyzed (Participants) | 50 | 24
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 7 | 3
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 13 | 9
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 16 | 11
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 3 | 4
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 800 | 392
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 8 | 4
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 17 | 8
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 11 | 5
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 4 | 0
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 697 | 324
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 3 | 4
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 6 | 5
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 9 | 5
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 3 | 4
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 614 | 232
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 4 | 2
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 6 | 4
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 9 | 4
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 3 | 0
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 514 | 183
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 5 | 2
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 7 | 3
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 4 | 2
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 5 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 413 | 140
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 2 | 2
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 5 | 0
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 3 | 3
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 3 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 352 | 90
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 0 | 1
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 5 | 1
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 2 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 2 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 266 | 71
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 1 | 0
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 1 | 0
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 1 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 1 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 188 | 41
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 1 | 0
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 0 | 0
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 1 | 1
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 114 | 20
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 1 | 0
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 1 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 0 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 38 | 8
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 0 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 6 | 1

39. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 53
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 53 are reported. Question 53 was following: "Did you have difficulty getting or maintaining an erection?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 50 | 24
  Baseline: not at all | 6 | 4
  Baseline: a little: number analyzed (Participants) | 50 | 24
  Baseline: a little | 19 | 5
  Baseline: quite a bit: number analyzed (Participants) | 50 | 24
  Baseline: quite a bit | 4 | 4
  Baseline: very much: number analyzed (Participants) | 50 | 24
  Baseline: very much | 21 | 11
  Baseline: not answered: number analyzed (Participants) | 50 | 24
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 10 | 8
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 8 | 8
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 8 | 4
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 13 | 7
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 800 | 392
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 6 | 2
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 8 | 6
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 8 | 3
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 18 | 6
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 697 | 324
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 4 | 6
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 6 | 5
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 0 | 1
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 11 | 6
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 614 | 232
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 3 | 1
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 4 | 4
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 4 | 2
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 11 | 3
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 514 | 183
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 7 | 3
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 2 | 2
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 3 | 2
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 9 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 413 | 140
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 2 | 1
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 5 | 1
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 1 | 1
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 5 | 2
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 352 | 90
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 1 | 0
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 3 | 1
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 1 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 4 | 1
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 266 | 71
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 0 | 0
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 1 | 0
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 0 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 3 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 188 | 41
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 1 | 0
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 0 | 1
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 0 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 1 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 114 | 20
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 1 | 0
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 0 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 38 | 8
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 0 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 6 | 1

40. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 54
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 54 are reported. Question 54 was following: "Did you have ejaculation problems (e.g, dry ejaculation)?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 50 | 24
  Baseline: not at all | 11 | 7
  Baseline: a little: number analyzed (Participants) | 50 | 24
  Baseline: a little | 14 | 4
  Baseline: quite a bit: number analyzed (Participants) | 50 | 24
  Baseline: quite a bit | 3 | 2
  Baseline: very much: number analyzed (Participants) | 50 | 24
  Baseline: very much | 22 | 11
  Baseline: not answered: number analyzed (Participants) | 50 | 24
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 13 | 11
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 5 | 5
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 3 | 1
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 18 | 10
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 800 | 392
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 12 | 10
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 9 | 1
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 5 | 0
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 14 | 6
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 697 | 324
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 7 | 6
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 3 | 5
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 1 | 1
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 10 | 6
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 614 | 232
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 8 | 3
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 2 | 1
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 1 | 2
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 11 | 4
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 514 | 183
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 7 | 4
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 0 | 0
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 3 | 0
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 11 | 4
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 413 | 140
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 5 | 2
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 3 | 0
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 0 | 1
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 5 | 2
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 352 | 90
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 3 | 2
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 1 | 0
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 0 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 5 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 266 | 71
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 1 | 0
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 0 | 0
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 0 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 3 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 188 | 41
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 2 | 0
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 0 | 1
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 0 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 114 | 20
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 1 | 0
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 0 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 38 | 8
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 0 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 6 | 1

41. Secondary Outcome: Number of Participants With European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Module Score for Question 55
Description: The EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It consisted of 25 questions (Question 31 to 55) distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions using 4 point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Number of participants with various responses to the question 55 are reported. Question 55 was following: "Have you felt uncomfortable about being sexually intimate?"
Time Frame: Baseline, Weeks 17, 33, 49, 65, 81, 97, 113, 129, 145,161 and 177
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 933 | 468
Participants
  Baseline: not at all: number analyzed (Participants) | 50 | 24
  Baseline: not at all | 31 | 13
  Baseline: a little: number analyzed (Participants) | 50 | 24
  Baseline: a little | 13 | 8
  Baseline: quite a bit: number analyzed (Participants) | 50 | 24
  Baseline: quite a bit | 4 | 0
  Baseline: very much: number analyzed (Participants) | 50 | 24
  Baseline: very much | 2 | 3
  Baseline: not answered: number analyzed (Participants) | 50 | 24
  Baseline: not answered | 0 | 0
  Week 17: not at all: number analyzed (Participants) | 839 | 419
  Week 17: not at all | 23 | 14
  Week 17: a little: number analyzed (Participants) | 839 | 419
  Week 17: a little | 11 | 7
  Week 17: quite a bit: number analyzed (Participants) | 839 | 419
  Week 17: quite a bit | 2 | 3
  Week 17: very much: number analyzed (Participants) | 839 | 419
  Week 17: very much | 3 | 3
  Week 17: not answered: number analyzed (Participants) | 839 | 419
  Week 17: not answered | 800 | 392
  Week 33: not at all: number analyzed (Participants) | 737 | 341
  Week 33: not at all | 24 | 10
  Week 33: a little: number analyzed (Participants) | 737 | 341
  Week 33: a little | 6 | 4
  Week 33: quite a bit: number analyzed (Participants) | 737 | 341
  Week 33: quite a bit | 6 | 2
  Week 33: very much: number analyzed (Participants) | 737 | 341
  Week 33: very much | 4 | 1
  Week 33: not answered: number analyzed (Participants) | 737 | 341
  Week 33: not answered | 697 | 324
  Week 49: not at all: number analyzed (Participants) | 635 | 250
  Week 49: not at all | 16 | 10
  Week 49: a little: number analyzed (Participants) | 635 | 250
  Week 49: a little | 4 | 6
  Week 49: quite a bit: number analyzed (Participants) | 635 | 250
  Week 49: quite a bit | 1 | 1
  Week 49: very much: number analyzed (Participants) | 635 | 250
  Week 49: very much | 0 | 1
  Week 49: not answered: number analyzed (Participants) | 635 | 250
  Week 49: not answered | 614 | 232
  Week 65: not at all: number analyzed (Participants) | 536 | 193
  Week 65: not at all | 13 | 5
  Week 65: a little: number analyzed (Participants) | 536 | 193
  Week 65: a little | 7 | 3
  Week 65: quite a bit: number analyzed (Participants) | 536 | 193
  Week 65: quite a bit | 1 | 2
  Week 65: very much: number analyzed (Participants) | 536 | 193
  Week 65: very much | 1 | 0
  Week 65: not answered: number analyzed (Participants) | 536 | 193
  Week 65: not answered | 514 | 183
  Week 81: not at all: number analyzed (Participants) | 434 | 148
  Week 81: not at all | 13 | 5
  Week 81: a little: number analyzed (Participants) | 434 | 148
  Week 81: a little | 6 | 1
  Week 81: quite a bit: number analyzed (Participants) | 434 | 148
  Week 81: quite a bit | 1 | 1
  Week 81: very much: number analyzed (Participants) | 434 | 148
  Week 81: very much | 1 | 1
  Week 81: not answered: number analyzed (Participants) | 434 | 148
  Week 81: not answered | 413 | 140
  Week 97: not at all: number analyzed (Participants) | 365 | 95
  Week 97: not at all | 8 | 3
  Week 97: a little: number analyzed (Participants) | 365 | 95
  Week 97: a little | 3 | 2
  Week 97: quite a bit: number analyzed (Participants) | 365 | 95
  Week 97: quite a bit | 1 | 0
  Week 97: very much: number analyzed (Participants) | 365 | 95
  Week 97: very much | 1 | 0
  Week 97: not answered: number analyzed (Participants) | 365 | 95
  Week 97: not answered | 352 | 90
  Week 113: not at all: number analyzed (Participants) | 275 | 73
  Week 113: not at all | 7 | 2
  Week 113: a little: number analyzed (Participants) | 275 | 73
  Week 113: a little | 0 | 0
  Week 113: quite a bit: number analyzed (Participants) | 275 | 73
  Week 113: quite a bit | 1 | 0
  Week 113: very much: number analyzed (Participants) | 275 | 73
  Week 113: very much | 1 | 0
  Week 113: not answered: number analyzed (Participants) | 275 | 73
  Week 113: not answered | 266 | 71
  Week 129: not at all: number analyzed (Participants) | 192 | 41
  Week 129: not at all | 3 | 0
  Week 129: a little: number analyzed (Participants) | 192 | 41
  Week 129: a little | 0 | 0
  Week 129: quite a bit: number analyzed (Participants) | 192 | 41
  Week 129: quite a bit | 1 | 0
  Week 129: very much: number analyzed (Participants) | 192 | 41
  Week 129: very much | 0 | 0
  Week 129: not answered: number analyzed (Participants) | 192 | 41
  Week 129: not answered | 188 | 41
  Week 145: not at all: number analyzed (Participants) | 116 | 21
  Week 145: not at all | 2 | 1
  Week 145: a little: number analyzed (Participants) | 116 | 21
  Week 145: a little | 0 | 0
  Week 145: quite a bit: number analyzed (Participants) | 116 | 21
  Week 145: quite a bit | 0 | 0
  Week 145: very much: number analyzed (Participants) | 116 | 21
  Week 145: very much | 0 | 0
  Week 145: not answered: number analyzed (Participants) | 116 | 21
  Week 145: not answered | 114 | 20
  Week 161: not at all: number analyzed (Participants) | 40 | 8
  Week 161: not at all | 1 | 0
  Week 161: a little: number analyzed (Participants) | 40 | 8
  Week 161: a little | 0 | 0
  Week 161: quite a bit: number analyzed (Participants) | 40 | 8
  Week 161: quite a bit | 1 | 0
  Week 161: very much: number analyzed (Participants) | 40 | 8
  Week 161: very much | 0 | 0
  Week 161: not answered: number analyzed (Participants) | 40 | 8
  Week 161: not answered | 38 | 8
  Week 177: not at all: number analyzed (Participants) | 6 | 1
  Week 177: not at all | 0 | 0
  Week 177: a little: number analyzed (Participants) | 6 | 1
  Week 177: a little | 0 | 0
  Week 177: quite a bit: number analyzed (Participants) | 6 | 1
  Week 177: quite a bit | 0 | 0
  Week 177: very much: number analyzed (Participants) | 6 | 1
  Week 177: very much | 0 | 0
  Week 177: not answered: number analyzed (Participants) | 6 | 1
  Week 177: not answered | 6 | 1

42. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment-emergent AE (TEAE) was defined as an AE that occurred from the date and time of the first dose of study drug through the date of last dose +30 days (or the day before initiation of a new antineoplastic treatment, whichever occurred first). AEs included both non-serious adverse events (AEs) and SAEs.
Time Frame: From first dose of study drug to the last dose + 30 days (or the day before initiation of a new antineoplastic treatment, whichever occurred first) (until the data cut-off date of 28 June 2017, maximum duration of treatment: 42.8 months)
Population: The safety population was defined as all participants randomly assigned to receive at least 1 dose or partial dose of study drug (enzalutamide or placebo) according to the actual treatment received (not the treatment assigned).
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 930 | 465
Participants
  AEs | 808 | 360
  SAEs | 226 | 85

43. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events Greater Than or Equal to Grade 3, Based on National Cancer Institute (NCI) Common Terminology Criteria (CTC) for AEs (CTCAE), Version 4.0
Description: An AE is any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. As per NCI CTCAE, Grade 3 events =medically significant but not immediately life-threatening, unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment, Grade 4 events =participant to be in imminent danger of death. Grade 5 events =death. A treatment-emergent AE (TEAE) was defined as an AE that occurred from the date and time of the first dose of study drug through the date of last dose +30 days (or the day before initiation of a new antineoplastic treatment, whichever occurred first).Number of participants with AEs of any of the Grade 3 or above (Grade 4, 5) were reported.
Time Frame: as for outcome 42
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 930 | 465
Participants | 292 | 109

44. Secondary Outcome: Number of Participants With Discontinuations From Study Treatment Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both non-serious adverse events (AEs) and SAEs.
Time Frame: as for outcome 42
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 930 | 465
Participants | 87 | 28

45. Secondary Outcome: Number of Participants With Increase of 2 or More National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) (Version 4.0) Toxicity Grades Above Baseline - Hematology
Description: Hematology parameters: Haemoglobin (grams per liter [g/L]); leukocytes (log 10 raised to power 9 per liter [10*9/L]); lymphocytes (log 10 raised to power 6 per liter [10*6/L]); neutrophils (log 10 raised to power 6 per liter [10*6/L]); platelets (log 10 raised to power 9 per litre [10*9/L]).
Time Frame: as for outcome 42
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 930 | 465
Participants
  Haemoglobin (Low) | 12 | 7
  Leukocytes (Low) | 7 | 7
  Lymphocytes (High) | 4 | 2
  Lymphocytes (Low) | 44 | 26
  Neutrophils (Low) | 13 | 4
  Platelets (Low) | 3 | 2

46. Secondary Outcome: Number of Participants With Increase of 2 or More National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) (Version 4.0) Toxicity Grades Above Baseline - Chemistry
Description: Chemistry parameters: Alanine aminotransferase (units per liter [U/L]); albumin (g/L); alkaline phosphatase (U/L); bilirubin (micromoles per liter [umol/L]); calcium (millimoles per liter [mmol/L]); creatine kinase (U/L); creatinine (umol/L); glucose, magnesium, phosphate, potassium, sodium (mmol/L).
Time Frame: as for outcome 42
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 930 | 465
Participants
  Alanine Aminotransferase (High) | 4 | 1
  Albumin (Low) | 7 | 0
  Alkaline Phosphatase (High) | 3 | 6
  Aspartate Aminotransferase (High) | 3 | 1
  Bilirubin (High) | 4 | 1
  Calcium (High) | 1 | 1
  Calcium (Low) | 2 | 1
  Creatine Kinase (High) | 4 | 3
  Creatinine (High) | 1 | 7
  Glucose (High) | 26 | 8
  Glucose (Low) | 5 | 1
  Magnesium (High) | 1 | 0
  Magnesium (Low) | 1 | 0
  Phosphate (Low) | 30 | 13
  Potassium (High) | 14 | 5
  Potassium (Low) | 0 | 3
  Sodium (High) | 2 | 1
  Sodium (Low) | 12 | 7

47. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs included Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and heart rate.
Time Frame: as for outcome 42
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide 160 mg | Placebo
Number analyzed (Participants) | 930 | 465
Participants
  SBP | 738 | 328
  DBP | 563 | 229
  Heart rate | 7 | 4

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug or till death, whichever occurred first (up to a maximum duration of 69.8 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Data reported in this section was collected and analyzed only for participants who were treated with at least 1 dose of study drug.
Groups:
- Placebo Patients Crossover to Enzalutamide 160 mg: Participants who received placebo in double-blind phase and who agreed to proceed to open-label phase, received 4 capsules of Enzalutamide 40 mg each (total dose of 160 mg per day), orally once daily (up to a maximum of 18.8 months) until radiographic progression. Participants after last dose of study drug, were followed up for safety up to 30 days and were long term followed up (for survival status and new prostate cancer therapies) to the death date or last known survival date.
Arm/Group | Enzalutamide 160 mg | Placebo | Placebo Patients Crossover to Enzalutamide 160 mg
All-Cause Mortality (participants affected / at risk) | 285/930 | 173/465 | 4/87
Serious Adverse Events (participants affected / at risk) | 372/930 | 100/465 | 12/87
Other Adverse Events (participants affected / at risk) | 762/930 | 299/465 | 45/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide 160 mg (N=930) | Placebo (N=465) | Placebo Patients Crossover to Enzalutamide 160 mg (N=87)
Anaemia (Blood and lymphatic system disorders) | 10 | 1 | 1
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 6 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 10 | 2 | 1
Angina pectoris (Cardiac disorders) | 3 | 0 | 0
Angina unstable (Cardiac disorders) | 3 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 9 | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 10 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 8 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 10 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 2 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 0
Chest pain (General disorders) | 7 | 1 | 0
Death (General disorders) | 2 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 3 | 0 | 1
Fatigue (General disorders) | 4 | 1 | 0
General physical health deterioration (General disorders) | 3 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0
Pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 3 | 2 | 0
Stent-graft endoleak (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 3 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 4 | 3 | 0
Intestinal congestion (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 2 | 0 | 0
Iodine allergy (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 6 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 3 | 0 | 0
Pneumonia (Infections and infestations) | 20 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Septic shock (Infections and infestations) | 3 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 2 | 0 | 0
Small intestine gangrene (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 11 | 6 | 0
Urosepsis (Infections and infestations) | 9 | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 12 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 5 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 4 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Venous injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | 0
Cerebral infarction (Nervous system disorders) | 4 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 7 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Diplegia (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 6 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 3 | 0 | 0
Spinal cord compression (Nervous system disorders) | 3 | 1 | 0
Syncope (Nervous system disorders) | 7 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 5 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0
Bladder hypertrophy (Renal and urinary disorders) | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 2 | 0
Calculus bladder (Renal and urinary disorders) | 2 | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 3 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 31 | 15 | 1
Hydronephrosis (Renal and urinary disorders) | 5 | 3 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 5 | 2 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 3 | 0
Postrenal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 2 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 7 | 8 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 2 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 2 | 2 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 3 | 0
Urinary fistula (Renal and urinary disorders) | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 3 | 1 | 0
Urinary retention (Renal and urinary disorders) | 13 | 12 | 0
Urinary tract obstruction (Renal and urinary disorders) | 4 | 2 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Bladder calculus removal (Surgical and medical procedures) | 1 | 0 | 0
Cystoprostatectomy (Surgical and medical procedures) | 1 | 0 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 4 | 0 | 0
Aortic dissection (Vascular disorders) | 2 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0
Haemorrhage (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 5 | 0 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Cardiac aneurysm (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Sinus arrest (Cardiac disorders) | 1 | 0 | 0
Tricuspid valve disease (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Performance status decreased (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 6 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Nail bed infection (Infections and infestations) | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chemical cystitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Vertigo CNS origin (Nervous system disorders) | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angiopathy (Vascular disorders) | 1 | 0 | 0
Aortic rupture (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide 160 mg (N=930) | Placebo (N=465) | Placebo Patients Crossover to Enzalutamide 160 mg (N=87)
Asthenia (General disorders) | 94 | 32 | 10
Fatigue (General disorders) | 348 | 73 | 13
Constipation (Gastrointestinal disorders) | 121 | 39 | 1
Diarrhoea (Gastrointestinal disorders) | 112 | 47 | 3
Nausea (Gastrointestinal disorders) | 125 | 42 | 3
Urinary tract infection (Infections and infestations) | 70 | 33 | 1
Fall (Injury, poisoning and procedural complications) | 164 | 25 | 2
Weight decreased (Investigations) | 80 | 11 | 4
Decreased appetite (Metabolism and nutrition disorders) | 108 | 22 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 119 | 36 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 120 | 38 | 4
Dizziness (Nervous system disorders) | 112 | 27 | 6
Headache (Nervous system disorders) | 103 | 23 | 3
Haematuria (Renal and urinary disorders) | 97 | 41 | 2
Urinary retention (Renal and urinary disorders) | 43 | 36 | 0
Hot flush (Vascular disorders) | 132 | 38 | 3
Hypertension (Vascular disorders) | 161 | 27 | 6
Anaemia (Blood and lymphatic system disorders) | 63 | 20 | 7
Oedema peripheral (General disorders) | 59 | 23 | 4
Rib fracture (Injury, poisoning and procedural complications) | 64 | 7 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 61 | 15 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 56 | 15 | 2
Pollakiuria (Renal and urinary disorders) | 43 | 25 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 15 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT02003924/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT02003924/SAP_003.pdf